

# NON-INTERVENTIONAL (NI) STUDY PROTOCOL

# **Study Information**

| Tenus. | 100 100 100 1 |
|---|---|
| Title | Effectiveness and Safety of Oral<br>Anticoagulants Among Obese Patients with<br>Non-Valvular Atrial Fibrillation in the<br>Veterans Affairs Population with Medicare |
| Protocol number | B0661162 |
| Protocol version identifier | 1.0 |
| Date | September 14, 2020 |
| Active substance | N/A |
| Medicinal product | Apixaban |
| Research question and objectives | The primary analysis will compare apixaban vs warfarin only. |
| | Primary Objectives: |
| | Aim 1: Evaluate the demographics and clinical characteristics of obese and severely obese NVAF patients initiating OACs (all patients, standard dose, and low dose). |
| | Aim 2: Determine if there is a difference in OAC treatment effect between obese and non-obese and severely obese and non-severely obese patients for stroke/systolic embolism (SE), MB, and net clinical benefit. |
| | Aim 3: Compare the risk of stroke/SE, major bleeding, net clinical benefit among obese and severely obese NVAF patients initiating OACs. |



This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# 1. TABLE OF CONTENTS 2. LIST OF ABBREVIATIONS......5 7. RATIONALE AND BACKGROUND......11 8. RESEARCH QUESTION AND OBJECTIVES ......12 9.2.2. Exclusion Criteria 16 9.4. Data Sources. 22 9.4.1. VA Database 23 9.7.2. Analysis Plan for Secondary CC

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | adverse event |
| AF | atrial fibrillation |
| ARIC | Atherosclerosis Risk in Communities |
| BMI | body mass index |
| CCI | ood, mass massi |
| CHADS <sub>2</sub> | Acronym: congestive heart failure, hypertension, age 75 years or older, diabetes mellitus |
| CMS | Center of Medicare Services |
| CPI | Consumer Price Index |
| CPT | Current Procedural Terminology |
| CrCl | creatinine clearance rate |
| DME | durable medical equipment |
| DOAC | direct aral anticoagulant |
| DSS | Decision Support System |
| EDB | enrollment database |
| ER | emergency room |
| GHP | group health plan |
| GLM | generalized linear models |
| GPP | Good Pharmacoepidemiology Practices |
| HAS-BLED | Hypertension, Abnormal Renal/Liver Function, Stroke, Bleeding, Labile INR, Elderly (Age >65 years), Drugs or Alcohol |
| HCFA | Health Care Financing Agency |
| HCPCS | Healthcare Common Procedure Coding System |
| HCRU | Healthcare resource utilization |
| HHA | Home Health Agency |
| HR | hazard ratios |
| ICD-9-CM | International Classification of Disease, Nineth Revision, Clinical Modification |
| ICD-10-CM | International Classification of Disease, Tenth Revision, Clinical<br>Modification |
| ICH | intracranial hemorrhage |
| IPTW | inverse probability treatment weightings |
| INR | international normalized ratio |
| LAB | laboratory |
| LAR | labartory results |
| LOS | length of stay |
| MB | major bleeding |
| NDE | non-destructive examinations |
| NVAF | non-valvular atrial fibrillation |
| OAC | oral anticoagulant |

| Abbreviation | Definition |
|--------------|----------------------------|
| PHA | pharmacy |
| PPPM | per patient per month |
| RAD | radiology |
| RIF | research identifiable file |
| RWD | real world data |
| SE | systolic embolism |
| SNF | skilled nursking facility |
| SSN | social security number |
| TTR | time in therapeutic range |
| USD | United States dollar |
| VA | Veterans' Affairs |
| VHA | Veterans' Health Affairs |
| VKA | Vitamin K antagonist |

# 3. RESPONSIBLE PARTIES

# Principal Investigator(s) of the Protocol

| Name, degree(s) | Title | Affiliation | Address |
|-----------------|---------|--------------------|-------------|
| PPD | PPD | Pfizer, Inc | Pfizer, NYC |
| PPD | PPD | PPD | PPD |
| PPD | PPD | BMS | PPD |
| PPD | PPD | Pfizer, Inc | Pfizer, NYC |
| PPD | PPD | PPD | PPD |
| PPD | PPD | Pfizer, Inc | Pfizer, NYC |
| PPD | PPD | PPD | PPD |
| PPD | PPD | Pfizer, Inc | Pfizer, NYC |
| PPD | PPD | STATinMED Research | PPD |
| PPD | Manager | STATinMED Research | PPD |
| PPD | Manager | STATinMED Research | PPD |

#### 4. ABSTRACT

**Title:** Effectiveness and Safety of Oral Anticoagulants Among Obese Patients with Non Valvular Atrial Fibrillation in the Veterans Affairs Population with Medicare

Rationale and Background: Prior RWD studies have evaluated the use of oral anticoagulants (OAC) in obese patients with atrial fibrillation (AF), but they are limited by sample size or by using ICD-9 diagnosis codes to define obesity. Conducting analyses of different datasets and addressing some of these limitations could add important information about the use of OACs in this population.

Research Question and Objectives: The overall objective of this analysis is to understand patient characteristics, use of treatment, and clinical outcomes among obese and severely obese patients with non-valvular atrial fibrillation (NVAF) who initiate therapy with OACs. The aim of this study is to compare all DOACs to warfarin; however, the primary analysis will be conducted among apixaban vs warfarin patients only. If sample size permits, we will also conduct other DOAC vs warfarin and DOAC vs DOAC analysis.

Study Design: This retrospective observational study will be conducted using linked national patient-level data from the Veterans Affairs (VA) Population and Center for Medicare and Medicare Services (CMS) fee-for-service database. The study period will be from January 1, 2013 through December 31, 2017. The study allows for a 6-month baseline period prior to the index date in the identification period. The index date will be defined as the date of first prescription for an OAC from July 1, 2013 − December 31, 2017; the first direct oral anticoagulant (DOAC) pharmacy claim date during the identification period will be designated as the index date. The first warfarin prescription date will be designated as the index date for patients without any DOAC claim. Patients will be required to have ≥1 AF medical claim in any position in the inpatient or outpatient setting before or on the index therapy date. Patients will be followed from the day after the index date until the earliest of 30 days after the date of discontinuation, switch, death, end of study period, or end of continuous medical enrollment (Parts A and B).

**Population:** Obese or severely obese AF patients in the CMS Medicare and Veterans' Health Affairs (VHA) databases who were newly prescribed OACs between January 1, 2013 and December 31, 2017.

Variables: Demographic and clinical characteristics and clinical outcomes including stroke/systolic embolism (SE), major bleeding (MB), and net clinical benefit.

**Data Sources:** The study will be conducted using linked CMS Medicare fee-for-service databases and Veterans Health Affairs Database.

**Study Size:** All eligible patients available for analysis will be included.

Data Analysis: Means, medians, and standard deviations will be provided for continuous variables. Numbers and percentages will be provided for dichotomous and polychotomous variables. Bivariate comparisons of baseline characteristics and outcomes measures will be provided. The primary analysis will be conducted among apixaban vs warfarin patients only. Inverse probability treatment weighting (IPTW) will be used to balance patient characteristics when comparing outcomes among different cohorts (for primary and secondary analyses). Appropriate tests (eg, t-test, chi-square test) will be used based on the distribution of the measure. Kaplan-Meier survival curves will be generated to illustrate the time to first Stroke/SE, MB Event, and Net Clinical Benefit. The cumulative incidence rate for clinical outcomes will be calculated. Cox proportional hazard ratio models will be used to evaluate the risk of clinical outcomes. Time to therapeutic range (TTR) will be calculated using the Rosendaal method and will be computed using INR values among warfarin patients during the follow-up. TTR will be calculated based on the percentage of time a patient remained in therapeutic range evaluated during the entire follow-up period. Data analysis will be executed using statistical software SAS version 9.4 (Cary, NC).

# 5. AMENDMENTS AND UPDATES

None.

#### 6. MILESTONES

| Milestone | Planned Date |
|--------------------------------------|-----------------------|
| Completion of protocol development | Draft 1: 1 July 2020 |
| Protocol revisions | Final: 14 August 2020 |
| Start of data collection | 10 June 2020 |
| End of data collection | December 2020 |
| Completion of Descriptive Tables | October 2020 |
| Completion of Multivariate Analysis | November 2020 |
| Completion of Dose Subgroup Analysis | December 2020 |
| Final Study Report | December 2020 |

#### 7. RATIONALE AND BACKGROUND

Atrial fibrillation (AF) is recognized as the most common sustained cardiac arrhythmia in the United States and is associated with a near five-fold excess of stroke. The prevalence of AF was estimated at 5.1 million in 2010 and projected to be 9.3 million in 2030 in the United States with an annual increase of 3.6%. AF also bears substantial economic burden. The direct health care costs associated with AF were estimated at approximately \$6 billion annually.

Vitamin K antagonists (VKAs; ie, warfarin) have been the mainstay treatment for stroke prevention among AF patients, reducing stroke by approximately 60%. Over the past 25 years, VKA use has been expanded from preventing stroke in valvular disease-associated AF patients to patients with non-valvular AF (NVAF).

Warfarin therapy requires close monitoring of the international normalized ratio (INR). The INR range from 2.0 to 3.0 (therapeutic range) was proven to be efficient in stroke prevention among AF patients, and is recommended in the treatment of AF.<sup>5,6</sup> However, due to its limited therapeutic index and possible drug and food interactions, only about half of AF patients in the United States receive warfarin therapy as recommended.<sup>7</sup>

Over the last several years, direct oral anticoagulants (DOACs), including apixaban, dabigatran, edoxaban, and rivaroxaban, were approved in the United States for stroke prevention among NVAF patients. Clinical trials demonstrated that DOAC use has shown stroke risk reduction similar or superior to warfarin, and lower or similar rates of bleeding. 8-11 In the years since their approval, DOACs have been increasingly preferred over warfarin due to

the convenience of fewer routine monitoring visits, no requirements for dose adjustment, and limited dietary interactions.

Obesity, another prevalent health condition in the United States, had an age-adjusted prevalence of 39.8% in 2015-2016. In the Atherosclerosis Risk in Communities (ARIC) study, obese and overweight individuals accounted for 17.9% of all AF cases; Additionally, obese patients have a 49% increased risk of AF compared with non-obese patients. Obese patients have been included in RCTs of DOACs and these studies did not show different results by weight. However, the severely obese population (BMI 40) has a more limited representation in RCTs. With the current fixed-dose DOAC prescriptions, the clinical impact of anticoagulation on NVAF patients with obesity is expected to be similar, provided patients have optimum peak and trough levels of DOACs.

Real world data (RWD) examining the use of oral anticoagulants (OACs) in obese and severely obese patients is limited by sample size or by using ICD-9 diagnosis codes to define obesity, with most literature focusing on outcomes of AF regardless of intervention. ARISTOPHANES obesity subgroup analysis found that in obese patients, apixaban was associated with lower risk of stroke/systemic embolism (SE) and major bleeding (MB) compared to warfarin. Rivaroxaban was associated with lower risk of stroke/SE but similar risk of MB, whereas dabigatran was associated with lower risk of MB, but similar risk of stroke/SE compared to warfarin. The goal of this study is to evaluate the risk of stroke/SE, MB, and net clinical benefit among obese and severely obese OAC treated patients using VA linked Medicare databases. The results of this linked, retrospective claims analysis will provide unique insight into outcomes of OAC use in obese and severely obese patients as the VA database includes vital measures (BMI, body weight, height) and laboratory results (INR, TTR) in addition to typical health outcomes from Medicare claims data.

# 8. RESEARCH QUESTION AND OBJECTIVES

# 8.1. Study Obectives

The overall objective of this analysis is to understand patient characteristics, treatment effect, and clinical outcomes among obese and severely obese patients with NVAF who initiate therapy with OACs (all patients, standard dose, and low dose). The primary analysis will be conducted among apixaban vs warfarin patients only.

#### 8.1.1. Primary Objectives

**Aim 1:** Evaluate the demographics and clinical characteristics of obese and severely obese NVAF patients initiating OACs (all patients, standard dose, and low dose; primary analysis will compare apixaban vs warfarin).

**Aim 2:** Determine if there is a difference in OAC treatment effect between obese and non-obese and severely obese and non-severely obese patients for stroke/SE, MB, and net clinical benefit.

**Aim 3:** Compare the risk of stroke/SE, MB, net clinical benefit among obese and severely obese NVAF patients initiating OACs (primary analysis will compare apixaban vs warfarin).

# 8.1.2. Secondary Objectives

**Aim 4**: A secondary analysis will also evaluate the following among warfarin treated obese and severely obese patients:

- Distribution of international normalized ratio (INR; <2, 2-3, >3).
- Distribution of time in therapeutic range (TTR ≥65% [good] and TTR <65% [poor]).</li>
- Compare the baseline characteristics of patients with good vs poor TTR.



#### 9. RESEARCH METHODS

# 9.1. Study Design

## 9.1.1. Key Index Period Definitions

- **Study Period:** The study period will range from January 1, 2013 through December 31, 2017.
- Patient Identification Period: The identification period will range from July 1, 2013 until December 31, 2017, allowing for a 6-month baseline period prior to the index date.
- Baseline Period: The baseline period will be 6 months prior to, and on, the index date
- Follow-up Period: The follow-up period will be defined as the time period between
  the day after the index date and end of study period (December 31, 2017). Patients
  will be followed from the day after the index date to 30 days after the date of
  discontinuation, switch, death, end of study period, or end of continuous medical
  enrollment (Parts A & B), whichever is earlier.

### 9.1.2. Key Index Point Definitions

- Index Therapy Date: The index date will be defined as the date of first prescription
  for an OAC from July 1, 2013 December 31, 2017; the first DOAC pharmacy claim
  date during the identification period (July 1, 2013-December 31, 2017) will be
  designated as the index date. The first warfarin prescription date will be designated as
  the index date for patients without any DOAC claim.
- AF Diagnosis: Evidence of AF diagnosis must be present, as evidenced from 1 or more claims for AF in any position in the inpatient or outpatient setting, before or on the index therapy date.

# Study Design Figure (for Illustration Purposes, May Not Be Proportionate):

Figure 1. Study Design



## 9.2. Setting

Adult patients prescribed a DOAC or warfarin will be selected between July 1, 2013 and December 31, 2017. Patients will be required to have one or more AF diagnosis claim in any position before or on index date. Patients will be required to have health plan enrollment (Parts A and B) for 6 months prior to the index date to ensure availability of complete patient medical history.

#### Follow-up Period:

The follow-up period will be defined as the time period between the day after the index date and end of study period (December 31, 2017). Patients will be followed from the day after the index date to 30 days after the date of discontinuation, switch, death, end of study period, or end of continuous medical enrollment (Parts A & B), whichever is earlier.

To assess first stroke/SE event, patients will be censored at first stroke/SE occurring anytime during period on the drug or within 30 days from the last day of days' supply of treatment prescription, 30 days after date of discontinuation, switch, death, end of study or end of continuous medical enrollment (Parts A and B), whichever is earlier.

To assess first MB event, patients will be censored at first major bleeding occurring anytime during period on the drug or within 30 days from the last day of days' supply of treatment prescription, 30 days after date of discontinuation, switch, death, end of study or end of continuous medical enrollment (Parts A and B), whichever is earlier.

For patients with stroke/SE or MB event, net clinical benefit will be assessed by evaluating the first hospital claim for a stroke/SE or MB. The hospital claim can occur anytime during the period of drug use or within 30 days from the last day of supply of treatment prescription.

### Other Factors Affecting Censoring During Follow-up

#### Discontinuation

Discontinuation will be defined as no evidence of index OAC prescription for 30 days from the last day of days' supply of last filled prescription. The date of discontinuation will be the last day of days' supply of last filled prescription. The follow-up will be censored at 30 days after the index drug discontinuation date.

#### Switch

Atrial fibrillation patients that receive a prescription for an OAC (warfarin, apixaban, dabigatran, edoxaban, or rivaroxaban) other than the index drug prescription during the follow-up period will be considered switchers if this OAC prescription is within  $\pm 30$  days of last days' supply. The follow-up will be censored at the switching of the index drug.

#### 9.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- Obese or severely obese.
- Initiated an OAC from July 1, 2013 December 31, 2017; the first DOAC pharmacy
  claim date during the identification period will be designated as the index date. The
  first warfarin prescription date will be designated as the index date for patients
  without any DOAC claim.
- Individuals ≥18 years old as of the index date.
- Had 6 months continuous health plan enrollment with medical benefits (Parts A & B) for at least 6 months pre-index date (baseline period).

- At least 1 diagnosis of AF prior to or on index date, identified by any medical claim associated with an International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) code of 427.31 or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code of I480-I482, and I4891.
- Had body weight or BMI value reported within ±6 months of the index date.

#### 9.2.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

- Had medical claims indicating a diagnosis or procedure of rheumatic mitral valvular heart disease, heart valve replacement/transplant, venous thromboembolism, or transient AF 6 months prior to or on the index date.
- Had hip/knee replacement surgery within 6 weeks prior to or on the index date.
- Were pregnant during the study period.
- Had an OAC prescription during the 6 months pre-index date.
- Had follow-up time equal to 0 days.
- Had more than one OAC on the index date.

Flag: A flag will be created to evaluate the mechanical heart valve/mitral stenosis during the 6 months prior to or on the index date using narrow definition.

All codes for the selection criteria are detailed in Appendix Table 4.

#### 9.2.3. Cohorts

After applying the selection criteria, patients will be assigned to the following subgroups based on body weight and BMI measures:

- 1. Obese Patients: Patients with body mass index (BMI) ≥30 or body weight ≥100 kg within ±6 months from the index date.
- 2. Non-Obese Patients: Patients not categorized as obese patients i.e. BMI <30 or body weight <100 kg patients within ±6 months from the index date will be designated as non-obese patients.
- 3. <u>Severely Obese Patients:</u> Patients with BMI >40 or body weight >120 kg within ±6 months from the index date.

Non-Severely Obese Patients: Patients not categorized as Severely Obese
ie, BMI ≤40 or body weight ≤120 kg patients within ±6 months from the index date
will be designated as non-severely obese patients.<sup>24</sup>

For patients that have multiple body weights during  $\pm 6$  months from the index date, the body weight closest to the index date will be used. Also, BMI will be given a preference over body weight in identifying patients into the above categories.

For each of the proceeding subgroup, patients will be categorized into the following cohorts based on their index OAC:

- Apixaban Cohort;
- b. Dabigatran Cohort;
- e. Edoxaban Cohort;
- d. Rivaroxaban Cohort;
- e. Warfarin Cohort.

The descriptive analysis will also be conducted separately among patients with low and standard dose OACs, defined below in Section 9.3 Variables.

#### 9.3. Variables

Baseline variables during the 6 months prior to, and on, the index date will be measured. Baseline variables will be evaluated using codes in any position unless noted otherwise.

 Table 1.
 Baseline Demographic and Clinical Characteristic Variables

| Variable | Data Source(s) | Operational Definition |
|---|---|---|
| Age | Both VA and<br>Medicare | Age will be defined as of the index date and used to assign patients to age groups (eg, 18-54, 55-64, 65-74, 75-79, ≥80 years). |
| Sex | Both VA and<br>Medicare | A flag will be created for female beneficiaries and reported as a percentage. |
| US Geographic<br>Region | Both VA and<br>Medicare | The United States will be divided into 5 regions:<br>Northeast, South, Midwest, West, and Other. |
| Race | Both VA and<br>Medicare | Race will be identified and will be categorized as:<br>White, Black, Other, and unknown. |
| Year of index OAC | Both VA and<br>Medicare | A flag will be created for proportion of unique patients with index OAC identified in 2013, 2014, 2015, 2016, and 2017. |

| Variable | Data Source(s) | Operational Definition |
|---|---|---|
| Dose of Index DOAC | Both VA and<br>Medicare | -Standard dose (apixaban 5 mg, dabigatran 150 mg, and rivaroxaban 20 mg) based on dose of the initial prescription of DOAC; -lower dose (apixaban 2.5 mg, dabigatran 75 mg, |
| | | rivaroxaban 15 mg/10 mg) based on dose of the initial prescription of DOAC. |
| Body Weight | VA | Body weight will be obtained as continuous and categorical variables. The categories will be: ≤60 kg 61-99 kg, 100-119 kg, and ≥120 kg. If a patient has multiple values, the value closest to the index date will be used. |
| BMI | VA | Body Mass Index: Body mass index will be calculated as weight in kilograms divided by the square of height in meters. Mean, median, and standard deviation will be provided for the continuous variable. The categories will be <18.5, 18.5-24.9, 25-29.9, 30-39, and ≥40. If a patient has multiple values, the value closest to the index date will be used. |
| Creatinine<br>Clearance | VA | Creatinine Clearance: Creatinine clearance will be identified using LOINC codes (2160-0, 33914-3, 48642-3, 48643-1, 62238-1, 2164-2, 14682-9). A categorical variable for the glomerular filtration rate (GFR) will be created with the following cutoff points: <15 ml/min, 15-29 ml/min, 30-59 ml/min, 60-89 ml/min, and ≥90 ml/min. If a patient has multiple values, the value closest to the index date will be used. The creatinine clearance rate (CrCl) will be calculated based on serum creatinine for patients who only had serum creatinine information. <sup>25</sup> |
| INR | VA | International Normalized Ratio Test Results will be identified using Logical Observation Identifiers Names and Codes (LOINC; 34714-6, 38875-1, 46418-0, 52129-4, 5895-7, 5896-5, 61189-7, 6301-6, 72281-9) occurring anytime during the baseline period will be evaluated. |
| CHADS <sub>2</sub> Score | Both VA and<br>Medicare | CHADS <sub>2</sub> Score will be calculated according to the points algorithm outlined in Appendix Table 5. |

| Variable | Data Source(s) | Operational Definition |
|---|---|---|
| CHA2DS <sub>2</sub> -VASc<br>Score | Both VA and<br>Medicare | CHA2DS2-VASc score will be calculated according to the points algorithm outlined in Appendix Table 6. |
| HAS-BLED Score | Both VA and<br>Medicare | HAS-BLED score will be calculated according to the points algorithm outlined in Appendix Table 7. |
| Baseline Medication<br>Use | Both VA and<br>Medicare | A flag will be created for the following medications prescribed during the baseline period: angiotensin-converting enzyme inhibitors/ angiotensin-receptor blockers, aspirin, beta blocker statins, proton pump inhibitors, H2-receptor antagonists, antiplatelets, nonsteroidal anti-inflammatory drugs, inhibitors of warfarin, inducers of warfarin, dronedarone, digoxin, calcium channel blockers, renin angiotensin system antagonists, glucocorticoids, diuretics, metformin, sulfonylureas, thiazolidinedione, insulin, other diabetes drugs, antiulcer agents, and antidepressant (See Appendix Table 8 for codes). |
| Bariatric Surgery | Both VA and<br>Medicare | A flag will be created for patients with claims for bariatric surgery (See Appendix Table 9 for codes). |
| CCI | Both VA and<br>Medicare | Charlson Comorbidity index will be calculated as a continuous variable (See Appendix Table 10 for calculation and codes). |
| Comorbid<br>Conditions | Both VA and<br>Medicare | The following comorbid conditions will be flagged in baseline: History of stroke/SE, history of bleeding, myocardial infarction, renal disease, liver disease, dyspepsia or stomach discomfort, diabetes, hypertension, congestive heart failure, non-stroke/SE peripheral vascular disease, anemia and coagulation defects, transient ischemic attack, coronary artery disease, peripheral artery disease (See Appendix Table 11 for codes). |

Table 2. Clinical and Outcome Variables

| Variable | Data<br>Source(s) | Operational Definition |
|---|---|---|
| Major Bleeding<br>Event | Both VA and<br>Medicare | Major bleeding event(s) observed during follow-up will be identified using hospital claims which had a MB diagnosis as the primary diagnosis code and occurring anytime during the follow-up period of drug use or within 30 days from the last day of supply of treatment prescription. A major bleeding event will be a dichotomous variable that equals 1 if there is ≥1 bleeding event during the follow-up period. Time to the first major bleeding event will be calculated. The first major bleeding event will be stratified by gastrointestinal (GI), intracranial hemorrhage (ICH), and other MB. (See Appendix Table 12 for codes). |
| Stroke/SE Event | Both VA and<br>Medicare | Stroke/SE will be identified using hospital claims which had a stroke/SE diagnosis code as the primary diagnosis code and occurring anytime during the period of drug use or within 30 days from the last day of supply of treatment prescription. Stroke/SE will be a dichotomous variable that equals 1 if there is ≥1 stroke event during the follow-up period. Time to the first stroke/SE event will be calculated. The first stroke/SE event will be stratified by ischemic stroke, hemorrhagic stroke, and SE. (See Append Table 12 for codes). |
| Net Clinical<br>Benefit | Both VA and<br>Medicare | For patients with stroke/SE OR MB event, net clinical benefit will be assessed by evaluating the first hospital claim for a stroke/SE or MB event. The hospital claim can occur anytime during the period of drug use or within 30 days from the last day of supply of treatment prescription. |
| INR | VA | International Normalized Ratio Test Results will be identified using Logical Observation Identifiers Names and Codes (LOINC; 34714-6, 38875-1, 46418-0, 52129-4, 5895-7, 5896-5, 61189-7, 6301-6, 72281-9) occurring anytime during the period of drug use or within 30 days from the last day of supply of treatment prescription. The mean |

| Variable | Data<br>Source(s) | Operational Definition |
|---|---|---|
| | | and median number of INR tests for warfarin patients will be calculated. The distribution of INR values (mean, median, maximum, minimum, Q1, Q3) will be evaluated descriptively and flags will be created for INR <2, 2-3, and >3. |
| Time in Therapeutic Range (TTR) | VA | TTR will be calculated using the Rosendaal method <sup>26</sup> and will be computed using INR values among warfarin patients during the follow-up. This method calculates INR-specific person-time by incorporating the frequency of INR measurements and their actual values, and assuming that changes between consecutive INR measurements are linear over time. TTR will be calculated based on the percentage of time a patient remained in therapeutic range evaluated during the entire follow-up period. Flags will be created for TTR ≥65% [good] and TTR <65% [poor]. |
| CCI | | |
| CCI | | |



#### 9.4. Data Sources

This retrospective observational study will be conducted using linked national patient-level data from the VA and Center for Medicare and Medicare Services (CMS) fee-for-service database and Veterans' Health Affairs database. The study period will be from January 1, 2013 through December 31, 2017. Patients with NVAF diagnosis will first be identified in VA dataset and then linked to Medicare data using social security number (SSN) as a unique patient identifier. Linked patient records will be deidentified before analysis. There will be no duplicate records and all outcomes will be counted only once in the linked database. Once the linked database is created, demographic, clinical, HRU, and cost outcomes will be available from the linked patient records using both Medicare and VA database. There will not be any overlapping HCRU or costs claims since VA is a closed system. If patient uses VA system then we will see a claim from VA database, if they use Medicare, they we will see a claim from Medicare database. So, all the claims will be unique with no overlapping.

In addition, VA data includes vital measures (BMI, body weight, height) and laboratory results (INR, TTR) that are not available in Medicare claims data. Using linked VA and Medicare data provides a more robust patient history as vital measures and laboratory results can be evaluated. BMI, body weight, and height are of importance when stratifying patients in obese and severely obese cohorts and INR and TTR allow evaluation of warfarin management. This study will add to an existing body of literature that evaluates various populations across different disease states the use linked VA and Medicare data to provide a more robust study population. <sup>27,28</sup>

Veterans' Health Affairs (VHA) Data

#### 9.4.1. VA Database

The VHA is the largest integrated health care system in the United States, providing care for veterans across the country. According to U.S. Department of Veterans Affairs (VA) estimates, there were approximately 24 million living veterans of the U.S. military in 2006. That year, the department provided medical services to more than five million of those veterans and to more than 400,000 other patients (ie, employees, eligible dependents and survivors of disabled veterans, and patients seen through sharing agreements with other providers such as the Department of Defense's TRICARE program). An additional 2.9 million veterans were enrolled in the system but did not seek services from the department that year, and the VA estimates that 5.8 million eligible veterans were never enrolled.<sup>29</sup>

The size and structure of the VHA system is quite different from most private care organizations. The system includes:

- 162 VA hospitals;
- 137 nursing homes;
- 43 domiciliaries;
- 850+ community and facility-based clinics;
- 14,800 doctors;
- 61,000 nurses; and
- 5 million patients.<sup>30</sup>

The system began as a network of hospitals and grew to include more aspects of care including clinics and nursing homes. Twenty-two regional networks, called the Veterans Integrated Service Networks (VISNs) have been created since 1995. Most VISNs consist of 7 to 10 hospitals, 25 to 30 ambulatory care clinics, 4 to 7 nursing homes, and 1 to 2 domiciliaries.<sup>31</sup>

The VHA Medical SAS® datasets are national administrative data for VHA-provided health care utilized primarily by veterans, but also by some non-veterans (eg, employees, research participants). The datasets are provided in SAS® format by fiscal year (FY) (October 1-September 30). These data are extracted from the National Patient Care Database (NPCD) as maintained by the VHA Office of Information at the Austin Information Technology Center (AITC), the central repository for VA data.

VHA Medical SAS® datasets include four inpatient datasets and two outpatient datasets. Variables common to both inpatient and outpatient data files include demographics (age, sex, race, birth date, marital status, city, county, and state of residence); period of military service; and selected special characteristics, including the patient's spinal cord injury status, prisoner of war history, and radiation or Agent Orange exposure. Also included are the patient's category of eligibility for VHA medical care, and the extent of a service-connected disability.

# VHA Medical SAS® Inpatient Datasets

The Medical SAS® Inpatient datasets cover four main categories of care: acute, extended, observation, and non-VA. Within each of these categories there are four datasets:

- Main: A patient's inpatient stay (episode of care);
- **Bed Section:** A patient's inpatient stay under a specified physician treating for a specialty service;
- Procedure: One day's procedure during an inpatient stay; and
- Surgery: One day's surgeries during an inpatient stay.

Inpatient variables describing each hospital admission include date, time, facility, and the primary diagnosis at admission. Discharge data include date, time, destination (eg, home, hospice, community nursing home), type of discharge (eg, regular, transfer to another hospital, death), and length of stay (LOS).

# VHA Medical SAS® Outpatient Datasets

Each outpatient data record represents one date of service for one outpatient, and includes a facility identifier, date and time of visit, and the type of clinic location where care was provided. Visits on a single day to multiple clinics, laboratories, and treatment programs are captured.

Outpatient care is reported in terms of diagnoses (International Classification of Diseases, 9<sup>th</sup> and 10<sup>th</sup> Revision, Clinical Modification [ICD-9-CM and ICD-10-CM] codes) and procedure (Current Procedural Terminology [CPT] codes), including dates and times. The type of provider for each service is reported using a VHA list of more than 500 categories (these may be changed in the future to agree with provider-type codes used by the Centers for Medicare and Medicaid Services [CMS]).

There currently are two Medical SAS® Datasets for outpatient care, visit and event.

- Visit: One day's occasions of service; and
- Event: One ambulatory encounter (coded as DSS Identifier/Clinic Stop).

### VHA Decision Support System

The VHA Decision Support System (DSS) is a managerial cost accounting system based on a commercial software named Eclipsys<sup>©</sup>. VHA modified Eclipsys<sup>©</sup> to interact with VistA and other VA national databases to populate the data elements required to allocate VHA costs to VHA products (goods and services provided during patient care). Introduced in 1994, full implementation of the VHA DSS in all facilities was completed in 1999.

The VHA DSS data files comprise a longitudinal, secondary relational database combining selected clinical data and fiscal (cost) data. The DSS provides a mechanism for integrating expenses, workload, and patient utilization. DSS information supports process and performance improvements by measuring quality of care, clinical outcomes, and financial impact. Within a fiscal year, periodic rollups of production data are performed to produce year-to-date non-destructive examinations (NDEs).

#### DSS Clinical NDEs

- Laboratory (LAB): Laboratory test utilization and costs (inpatient and outpatient);
- Laboratory Results (LAR): Laboratory test results for a specific list of tests (inpatient and outpatient);
- Pharmacy (PHA): Pharmacy prescription utilization and costs (inpatient and outpatient); and
- Radiology (RAD): Radiological procedure utilization and costs.

The stability of VHA data sources allows for superior analysis of the continuity of care of patients over multiple years.

#### US Centers for Medicare & Medicaid Services (CMS) Data

#### Medicare Inpatient Data

The inpatient claim file contains final action claims data submitted by inpatient hospital providers for reimbursement of facility costs. Some information contained in this file includes diagnosis (International Classification of Diseases, Ninth and Tenth Revision, Clinical Modification [ICD-9-CM and ICD-10-CM] diagnosis code, procedure (ICD-9 and ICD-10 procedure code), diagnosis-related group (DRG), dates of service, reimbursement amount, hospital provider, and beneficiary demographic information. Each observation in this file is at the claim level.

### Medicare Outpatient Data

The outpatient claim file contains final action claims data submitted by institutional outpatient providers. Examples of institutional outpatient providers include hospital outpatient departments, rural health clinics, renal dialysis facilities, outpatient rehabilitation facilities, comprehensive outpatient rehabilitation facilities, and community mental health centers. Some information contained in this file includes diagnosis and procedure (ICD-9-CM diagnosis, ICD-9 procedure, ICD-10 diagnosis, ICD-10 procedure, Centers for Medicare and Medicaid Service [CMS] Healthcare Common Procedure Coding System [HCPCS] codes), dates of service, reimbursement amount, outpatient provider number, revenue center codes, and beneficiary demographic information. Each observation in this file is at the claim level.

# Medicare Part D Drug Events (PDE) Data

The PDE data contains prescription drug costs and payment data (including out-of-pocket costs [co-payments and deductibles]) that enable CMS to make payments to the plans and otherwise administer Part D benefits. When a beneficiary fills a prescription under Medicare Part D, a prescription drug plan sponsor must submit a summary record to CMS. The PDE data are not the same as individual drug claim transactions but are summary extracts using CMS-defined standard fields.

Skilled Nursing Facility (SNF) Research Identifiable File (RIF)

The SNF file contains final action, fee-for-service (FFS) claims data submitted by SNF providers. This file includes ICD-9-CM and ICD-10-CM diagnosis and procedure codes, dates of service, reimbursement amount, SNF provider number, and beneficiary demographic information.

Home Health Agency (HHA) RIF

The HHA file contains final action, FFS claims submitted by HHA providers. This file includes: number of visits, type of visit (skilled nursing care, home health aides, physical therapy, speech therapy, occupational therapy, and medical social services), diagnosis (ICD-9-CM and ICD-10-CM diagnosis), date of visit, reimbursement amount, HHA provider number, and beneficiary demographic information.

#### Hospice RIF

The Hospice file contains final action claims submitted by hospice providers. Once a beneficiary elects hospice care, all hospice-related claims will be found in this file, regardless of if the beneficiary is in Medicare FFS or in a Medicare managed care plan. This file includes level of hospice care received (eg, routine home care, inpatient respite care), terminal diagnosis (ICD-9-CM and ICD-10-CM diagnosis), dates of service, reimbursement amounts, hospice provider number, and beneficiary demographic information.

# Durable Medical Equipment (DME) RIF

The DME file contains final action, FFS claims submitted by DME suppliers. This file includes diagnosis (ICD-9-CM and ICD-10-CM diagnosis), services provided (CMS Common Procedure Coding System [HCPCS] codes), dates of service, reimbursement amounts, DME provider number, and beneficiary demographic information.

#### Medicare Carrier File

The Carrier file (also known as the Physician/Supplier Part B claims file) contains final action, FFS claims submitted on a CMS-1500 claim form. Most of the claims are from non-institutional providers, such as physicians, physician assistants, clinical social workers, and nurse practitioners. Claims for other providers, such as free-standing facilities, are also found in the Carrier file. Examples include independent clinical laboratories, ambulance providers and free-standing ambulatory surgical centers. This file includes diagnosis and procedure codes, dates of service, reimbursement amounts, provider numbers, and patient demographic information.

#### Medicare Denominator File

The denominator file contains demographic and enrollment information of Medicare beneficiaries enrolled or entitled in a given year. It combines Medicare beneficiary entitlement status information from administrative enrollment records with third-party payer information and group health plan (GHP) enrollment information. It is an abbreviated version of the enrollment database (EDB) (selected data elements).

Some information contained in this file includes the beneficiary's unique identifiers, state and county codes, ZIP codes, dates of birth, dates of death, sex, race, age, monthly entitlement indicators (A/B/both), reasons for entitlement, state buy-in indicators, and monthly managed care indicators (yes/no). However, all Medicare files described above can be linked by de-identified patient ID and will be included in the same CMS access request.

Data are collected on an ongoing basis with files constructed annually. It does not contain data on all beneficiaries ever entitled to Medicare. The file contains data only for beneficiaries who were entitled during the year of the data. These data are available annually in May of the current year for the previous year.

#### 9.5. Study Size

All elibgile patients available for analysis will be included.

A feasibility analysis was conducted to examine the sample size of patients available in the linked VA and Medicare dataset with diagnosis of NVAF and BMI or body weight reported within  $\pm 6$  months of index diagnosis. Enrollment in Medicare Part D was removed as an inclusion criterion during the feasibility analysis as 50% of the study population would be excluded. Many patients in this study population use VA prescription drug benefits due to

cost savings over Medicare Part D. However, we will identify OAC use from Medicare Part D in patients who have this coverage along with VA pharmacy benefits. Approximately 56,000 patients would be included in this study population, with 20,000 included in the apixaban cohort. The VA feasibility study results and hazard ratios (HR) were used to calculate the needed sample size below.

A power calculation was completed for effectiveness outcomes comparing the difference between stroke rates using an alpha of 0.05, power of 80%, an accrual period of 4.5 years (identification period where patients are selected into the study), and a loss of follow-up of 55% for the warfarin cohort and 40% for the apixaban cohort. Using the stroke hazard ratio of 0.63 (from ARISTOPHANES Obesity subgroup<sup>23</sup> and an incidence rate of 1.10 per 100 person-years (from VA-Medicare feasibility analysis conducted in Q1-Q2 2020) in the warfarin group, a Cox proportional hazards analysis of stroke would need 7,945 patients per cohort (1:1 matching).

• Accrual Period: 4.5 years (identification period).

• Loss of follow-up: 55% for the warfarin cohort and 40% for the apixaban cohort.

Alpha: 0.05.

Power: 80%.

Table 3. Power Calculation

| Hazard Ratio (HR)<br>Apixaban vs Warfarin | | Incidence Rates for Stroke/SE<br>(per 100 person-years) | | Stroke/SE<br>Sample Size | | |
|---|---|---|---|---|---|---|
| HR | Source | Rate<br>(warfarin) | Source | Apixaban | Warfarin | Total |
| OBESI' | ГҮ | * | <del>5</del> 6 | <del>.</del> | | |
| 0.63 | ARISTOPHANES-<br>Obesity subgroup <sup>23</sup> | 1.80 | ARISTOPHANES-<br>Obesity subgroup | 4,882 | 4,882 | 9,764 |
| 0.63 | ARISTOPHANES-<br>Obesity subgroup | 1.10 | VA Feasibility | 7,945 | 7,945 | 15,890 |
| 0.76 | Sandhu et al <sup>19</sup> | 1.28 | Sandhu et al | 17,769 | 17,769 | 35,538 |
| 0.76 | Sandhu et al | 1.10 | VA Feasibility | 20,646 | 20,646 | 41,292 |
| SEVER | E OBESITY | | | 10. | | 200 |
| 0.72 | ARISTOPHANES-<br>Obesity subgroup | 1.60 | ARISTOPHANES-<br>Obesity subgroup | 10,195 | 10,195 | 20,390 |
| 0.72 | ARISTOPHANES-<br>Obesity subgroup | 0.87 | VA Feasibility | 18,640 | 18,640 | 37,280 |
| 0.39 | Hohnloser et al <sup>32</sup> | 1.13 | Hohnloser et al | 2,356 | 2,356 | 4,712 |
| 0.39 | Hohnloser et al | 0.87 | VA Feasibility | 3,055 | 3,055 | 6,110 |

Sandhu et al used BMI ≥30 kg/m²; Hohnloser et al used weight >120 kg

### 9.6. Data Management

N/A.

### 9.7. Data Analysis

All variables will be analyzed descriptively. Cohorts will be compared; however, the main analysis will be between apixaban vs warfarin. Other comparisons (DOAC vs warfarin and DOAC vs DOAC) will be optional depending on the sample size. Means, medians, and standard deviations will be provided for continuous variables when performing descriptive analysis of continuous data. Numbers and percentages will be provided for dichotomous and polychotomous variables when performing descriptive analysis of categorical data. Bivariate comparisons of baseline characteristics and outcomes measures will be provided. Appropriate tests (eg, t-test, chi-square test) will be used based on the distribution of the measure. The incidence rate of stroke/SE, MB, and net clinical benefit will be calculated. The incidence rate will be calculated as the number of patients who experience the event divided by the observed time at risk. Kaplan-Meier survival curves will be generated to illustrate time-to-first stroke/SE, MB, and net clinical benefit. Statistical tests of significance will be conducted to determine differences between the cohorts. Baseline and outcome tables will be stratified by obese, severely obese, and index dose of DOAC.

All data analysis will be executed using statistical software SAS version 9.4 (Cary, NC).

## 9.7.1. Analysis Plan for Primary Objective

Baseline demographic and clinical factors such as age, sex, geographic region, baseline medications, and co-morbidities among NVAF patients initiating OAC will be summarized. Descriptive statistics, (ie, mean, standard deviation, median, and inter-quartile range for continuous variables and differences across treatments) will be compared using the Student's t-test or Wilcoxon rank sum test. Percentages for categorical and binary variables will be presented for all baseline patient characteristics and will be compared using the chi-square test or Fisher's Exact test.

The cumulative incidence rate for clinical outcomes (stroke/SE, MB, net clinical benefit) will be calculated. MB will be stratified by GI bleeding, ICH, and other bleeding; Stroke/SE will be stratified by hemorrhagic, ischemic, and systemic embolism. The incidence rate will be calculated as the number of patients who experience the event divided by the observed time at risk. The incidence rate will be calculated per 100 person-years.

### Inverse Probability Treatment Weighting (IPTW)

Inverse probability treatment weighting (IPTW) will be used to balance patient characteristics when comparing outcomes among different cohorts. Three sets of IPTW will be conducted (all patients, obese patients, and severely obese patients). Depending on sample size, IPTW will also be conducted for the standard dose patients separately. In addition, the primary analysis will be conducted for apixaban vs warfarin and depending on the sample size, other OAC comparisons will be conducted.

IPTW uses propensity scores to obtain estimates of the average treatment effect. The propensity score will be calculated using a logistic model with treatment cohorts included in the model, using warfarin patients as the reference (ie, control cohort). The propensity score is defined as the probability of a patient receiving a certain treatment or not conditional on their observed baseline covariates (eg, age, gender, comorbidities, medications, etc.). The list of variables included in the logistic model will be based on clinical rationale. The propensity score acts as a balancing score between the cohorts. After calculating the propensity score, the distribution of the propensity scores will be reviewed. Each patient will be weighted by the inverse of the probability of their treatment option (weight=1/propensity score).

If a treated patient has a very low propensity score, a very large weight will be generated. Large weights can increase the variability of estimated treatment effect. In order to address this, the weights will be stabilized. In order to stabilize the weights, the treatment option and control weights will be multiplied by a constant, equal to the expected value of being in the treatment or comparison cohorts, respectively (see below). This reduces the variability of the weights and reduces the variance of the treatment effect estimates.

$$\frac{\sum_{i=1}^{N_T} PS_i}{N_T} * \frac{1}{PS_i}$$

The distribution of the stabilized weight will be reviewed. If no extreme outliers are observed, the stabilized weights will be applied to the sample. In cases of extreme outliers, the large weights could be set to a less extreme value (eg, recoding all weights that are outside 5<sup>th</sup> and 95<sup>th</sup> percentile to the 5<sup>th</sup> and 95<sup>th</sup> value, respectively). If needed, truncation can be done after stabilizing the weights.

After the weights are applied, the balance of the baseline covariates will be assessed. First, the means and proportions of baseline variables will be compared. The standardized difference compares the difference in means in units of the standard deviation. If the standardized difference is less than 10%, the covariates will be considered balanced. For continuous variables, the balance of the distribution will also be assessed. The high-order movements and interactions between variables should be similar between cohorts. The standardized difference will be used to compare the mean of the square of continuous variables. Graphical comparisons of the distribution of continuous variables will be completed. Side-by-side boxplots and empirical cumulative distribution functions will be used to the compare the distribution of continuous covariates in the unweighted and weighted samples. Since the graphical approach can be subjective, a numerical method for comparing the distribution of continuous baseline covariates will also be completed. Kolmogorov-Smirnov test allows a comparison of the distribution of a continuous variable between two independent groups. 33-36

# Cox Proportional Hazards Model

Cox models will be used to compare the risk of stroke/SE, MB, and net clinical benefit between cohorts. Variables that are not balanced in the weighted population will be included in the models in addition to treatment variables. For the secondary objective, an interaction term for treatment and obesity status will be included in the models. The proportional hazards assumption will be evaluated by visually inspecting the Kaplan-Meier plot. It the proportional hazards assumption appears to be violated, it will be confirmed by testing the significance of interactions between treatment and log of time.

# 9.7.2. Analysis Plan for Secondary CC

Any further comparisons or sub-group analysis will be assessed and conducted based on feasibility analysis to ensure adequate sample size through power calculation.



# Sensitivity Analysis: Propensity Score Matching

The propensity score matching (PSM) technique will be used to control for potential confounders when comparing the cohorts.<sup>37</sup> Covariates to be included in the logistic regression model may include the following variables: age, geographic region, Charlson comorbidity index score, comorbidities, and other clinical characteristics. The final list of

variables to be used in the model will be discussed and determined during analysis development, after reviewing the pre-matched descriptive tables. Each subject in the reference cohort will be matched to a subject in the comparator cohort with the closest propensity score. The nearest neighbor method without replacement and with a caliper of 0.01 will be used to select the matched samples. The balance of covariates between treatment groups will be determined using the absolute standardized difference of the mean ≤0.10.

After PSM, no significant differences are expected among all pre-index measures between the patient cohorts. PSM with a different ratio (1:2 or 1:3) can also be considered if the matched sample size using a ratio of 1:1 is too small.

### 9.8. Quality Control

STATinMED Research's approach combines scientific rigor with accurate results. The company focuses on quality at each step of the process, including, but not limited to the following:

- Sound scientific design and clinically rigorous review.
- Detailed study protocol, that includes definitions, codes, analyses, and table shells. A
  member of the STATinMED clinical team will review the appropriateness and
  validity of the coding strategy and identify relevant issues. The protocol further
  provides STATinMED Research and Pfizer the opportunity to solidify research
  questions and to address any potential gaps in information.
- Rigorous quality assurance checks will be performed during the construction of the
  dataset. Several checks are used, including record-level verification of all data
  elements, double programming of certain portions of the dataset, programming data
  edit checks, visual review of raw data against the constructed data elements, and
  review of analysis to assess validity of results.
- STATinMED Research's analysis will be performed by an analyst under the supervision of the project manager, lead analyst, and/or vice president. These team members review programs and output for consistency with the analysis plan, quality, and accuracy. Further, results will be reviewed with Pfizer to establish that the results meet Pfizer's expectations.

Additional quality control procedures are enlisted below.

| QC Checklist | Initials |
|---|---|
| QC of Excel File | |
| <ul> <li>Evaluate each step of attrition table (eg, check percentage drop at each step,<br/>compare to prior studies (rerun, other internal, external (if applicable)).</li> </ul> | |
| <ul> <li>5 separate database equal total pooled population (pre-match and post-match)</li> </ul> | ). |
| <ul> <li>Check percentage drop after PSM (expect ~10% drop but dependent on<br/>database/original sample size; add PSM sample size to attrition table).</li> </ul> | |
| <ul> <li>Baseline table → ensure all categorical variables equal 100% and total samplesize, make sure all three dose variables are complete (Auto-check using formulas).</li> </ul> | e |
| <ul> <li>Outcome table → components of MB or stroke/SE should be equal or larger<br/>than overall MB or stroke/SE (N and incidence rates; auto check using<br/>formula), all other categorical variables equal 100% and total sample size,<br/>minimum follow-up should be at least 1 day and check distribution.</li> </ul> | |
| <ul> <li>Outcome table → ensure incidence rates can be calculated using number of<br/>events and person time</li> </ul> | |
| <ul> <li>Check conditional formatting for p-values and standardized difference (red for p-values &lt;0.05 (unless interaction p-value where the cutoff is &lt;0.10), green for standardized difference ≥10.00).</li> </ul> | |
| <ul> <li>(Rerun) Compare percent difference between original and new results<br/>(10% cutoff) in baseline and outcome tables (using formula).</li> </ul> | |
| <ul> <li>Compare incidence rates, KM curves, and Cox model results to ensure<br/>alignment (eg, compare log rank test to Cox model, visually inspect KM curv<br/>can calculate IRR to see similarity to HR).</li> </ul> | /е, |
| <ul> <li>Ensure pooled dose pre-match table has the same sample size as indicated in<br/>baseline table.</li> </ul> | |
| <ul> <li>Sample size in subgroup matches the sample size in baseline table (eg, CHF subgroup tables match CHF baseline row in pooled baseline table). For each analysis, will be customized for the subgroups.</li> </ul> | |
| <ul> <li>Sample size of combined subgroup equals total population (for interaction).</li> </ul> | |
| <ul> <li>If lower CI is &gt;1 or upper CI is &lt;1, then p-value should be &lt;0.05 (using formula).</li> </ul> | |
| <ul> <li>Check duplicates within a sheet for Cox models (using formula).</li> </ul> | |
| Data Integrity Review Tasks for Publications (will be customized for each manuscript each figure and table will be listed) – Completion by medical writer and data check against excel file by non-project team member | 2 |
| Check whether all data sources are annotated and traceable for future retrieval. | |
| Check the following data by comparing it against the appropriate source documentation (including, but not limited to): | n |

| QC Checklist | Initials |
|---|---|
| QC of Excel File | |
| <ul> <li>Numbers, units, and symbols (for example, &gt;, &lt;, ≥, *) in text.</li> </ul> | |
| Numbers, units, and symbols in all tables. | |
| <ul> <li>Numbers and units (including those on axes) and symbols in all figures,<br/>including flow charts and diagrams.</li> </ul> | |
| Measurement units. | |
| Data-driven statements. | |
| Check that all data values are consistent throughout the document sections, tables, figures, legends, and footnotes (for example, data in the abstract match data in the body of document, and results section match figure). | |
| Check that values from other sources match reference. | |
| For any items not completed and marked N/A, provide rationale below. | |
| Additional comments. | |
| Click here to enter text. | |

#### 9.9. Limitations of the Research Methods

A key strength of this study design is that retrospective observational analyses provide a better understanding about the study population in real-world clinical practice and offer complimentary information to controlled clinical trials. Retrospective observational studies also allow the evaluation of patients who are often under-represented in clinical trials, such as those with comorbidities and older adults. Since prescribing patterns in the real world can be complex, retrospective analysis provides a more comprehensive picture of how medications are used by clinicians in routine practice. In addition, the claims databases include all medical and pharmacy claims of patients and allow for longitudinal analysis of a nationally representative sample.

A second key strength of this study design is the linked VA and Medicare databases, which allow us to see a comprehensive patient journey and health resource utilization across two databases. The VHA database includes lab values that will be used to identify obese and severely obese patients as opposed to ICD codes only. Additionally, INR values are available in the VHA data, which will also be evaluated to provide insights into warfarin management.

While claims data are extremely valuable for the efficient and effective examination of health care outcomes, treatment patterns, HCRU, and costs, all claims databases have certain inherent limitations because the claims are collected for administrative purposes and not research. For instance, the presence of a claim for a filled prescription does not indicate that the medication was taken as prescribed or at all. Medications filled over the counter or provided as samples by the physician cannot be observed in the claims data. And the presence of a diagnosis code on a medical claim does not indicate the positive presence of

disease, as the diagnosis code may be incorrectly coded or included as rule-out criteria rather than actual disease.

# 9.10. Other Aspects

Not Applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient Information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 10.2. Patient Consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

## 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

N/A.

# 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE).

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

In the event of any prohibition or restriction imposed (eg, clinical hold) by an applicable competent authority in any area of the world, or if the investigator is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

An Excel file will be provided with all the descriptive and multivariate analysis tables. A final study report detailing the final study protocol and the analysis results will be provided when the study is complete.
#### 13. REFERENCES

- Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: The Framingham Study. Stroke. 1991;22(8):983-8.
- Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the US adult population. Am J Cardiol. 2013;112(8):1142-7.
- 3. Roger VL, Go AS, Lloyd-Jones DM, et al. Heart disease and stroke statistics—2012 update a report from the American Heart Association. *Circulation*. 2012;125(1):e2-e220.
- 4. Hart RG, Pearce LA, Aguilar MI. Meta-analysis: Antithrombotic therapy to prevent stroke in patients who have non-valvular atrial fibrillation. *Ann Internal Med*. 2007;146(12):857-67.
- 5. Fuster V, Rydén LE, Asinger RW, et al. ACC/AHA/ESC guidelines for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines and Policy Conferences (Committee to Develop Guidelines for the Management of Patients With Atrial Fibrillation) Developed in collaboration with the North American Society of Pacing and Electrophysiology. J Am Coll Cardiol. 2001;38(4):1231-65.
- 6. Stroke Prevention in Atrial Fibrillation Investigators. Adjusted-dose warfarin versus low-intensity, fixed-dose warfarin plus aspirin for high-risk patients with atrial fibrillation: Stroke Prevention in atrial fibrillation III randomised clinical trial. *Lancet*. 1996;348(9028):633-8.
- 7. Harburger JM. Aronow WS. Newer anticoagulants for non-valvular atrial fibrillation. *Pharmaceuticals*. 2012;5(5):469-80.
- 8. Lip GYH, Halperin JL, Petersen P, Rodgers GM, Pall D, Renfurm RW. A phase II, double-blind, randomized, parallel group, dose-finding study of the safety and tolerability of darexaban compared with warfarin in patients with non-valvular atrial fibrillation: the oral factor Xa inhibitor for prophylaxis of stroke in atrial fibrillation study 2 (OPAL-2). *J Thrombrosis Haemostasis*. 2015;13:1405-13.
- 9. O'Donoghue ML, Ruff CT, Giugliano RP, et al. Edoxaban vs. warfarin in vitamin K antagonist experienced and naive patients with atrial fibrillation. *Eur Heart J.* 2015;36(23):1470-7.
- Agnelli G, Buller HR, Cohen A, et al. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013;368(8):699-708.

- Lanssen M, Raskob G, Gallus A, et al. Apixaban versus enoxaparin for thromboprophylaxis after knee replacement (ADVANCE-2): A randomized doubleblind trial. *Lancet*. 2010;375(9717):807-15.
- Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of obesity among adults and youth: United States, 2015-2016. NCHS Data Brief 2017;288:1-8.
- 13. Huxley RR, Lopez FL, Folsom AR, et al. Absolute and attributable risks of atrial fibrillation in relation to optimal and borderline risk factors. *Circulation*. 2011 April 12;123(14).
- Aromolaran AS, Boutjdir M. Cardiac ion channel regulation in obesity and the metabolic syndrome: relevance to long qt syndrome and atrial fibrillation. Front Physiol. 2017;8:431.
- 15. Ezekowitz ME, Parise H, Connolly SJ, et al. The use of dabigatran according to body mass index: the RE-LY experience. Eur Heart J 2014;35:1111.
- Connolly SJ, Ezekowitz MD, Yusuf S, et al. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med 2009;361:1139-51.
- 17. Balla SR, Cyr DD, Lokhnygina Y, et al. Relation of Risk of Stroke in Patients With Atrial Fibrillation to Body Mass Index (from Patients Treated With Rivaroxaban and Warfarin in the Rivaroxaban Once Daily Oral Direct Factor Xa Inhibition Compared with Vitamin K Antagonism for Prevention of Stroke and Embolism Trial in Atrial Fibrillation Trial). Am J Cardiol 2017;119:1989-96.
- 18. Granger CB, Alexander JH, McMurray JJ, et al. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med 2011;365:981-92.
- Sandhu RK, Ezekowitz J, Andersson U, et al. The 'obesity paradox' in atrial fibrillation: observations from the ARISTOTLE (Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation) trial. Eur Heart J 2016;37:2869-78.
- Boriani G, Ruff CT, Kuder JF, et al. Relationship between body mass index and outcomes in patients with atrial fibrillation treated with edoxaban or warfarin in the ENGAGE AF-TIMI 48 trial. Eur Heart J 2019;40:1541-50.
- Zukkoor, S. Expert Analysis: Antiarrhythmic and DOAC Dosing in Obesity. American College of Cardiology (2019). https://www.acc.org/latest-incardiology/articles/2019/07/03/08/22/antiarrhythmic-and-doac-dosing-in-obesity. Accessed June 2, 2020.
- Prioetti M, Guiducci E, Cheli P, Lip, G. Is There an Obesity Paradox for Outcomes in Atrial Fibrillation? A Systematic Review and Meta-Analysis of Non-Vitamin K Antagonist Oral Anticoagulant Trials. Stroke 2017;48(4):857-566.

- Deitelzweig, S., Keshishian, A., Kang, et al. (2020). Effectiveness and Safety of Oral Anticoagulants among NVAF Patients with Obesity: Insights from the ARISTOPHANES Study. Journal of Clinical Medicine, 9(6), 1633.
- 24. Centers for Disease Control and Prevention. Defining Adult Overweight and Obesity (2020). https://www.cdc.gov/obesity/adult/defining.html. Accessed June 26, 2020.
- CKD-EPI Creatinine Equation (2009). National Kidney Foundation. https://www.kidney.org/content/ckd-epi-creatinine-equation-2009. Accessed February 21, 2018.
- 26. Reiffel J. Time in the Therapeutic Range for Patients Taking Warfarin in Clinical Trials. *Circulation*. 2017;135:1475–1477. DOI: 10.1161/CIRCULATIONAHA.116.026854.
- Radomski TR, Zhao X, Thorpe CT, et al. VA and Medicare Utilization Among Dually Enrolled Veterans with Type 2 Diabetes: A Latent Class Analysis. *J Gen Intern Med* 2016;31(5):524-531.
- Wang V, Coffman CJ, Stechuchak KM, et al. Comparative Assessment of Utilization and Hospital Outcomes of Veterans Receiving VA and Non-VA Outpatient Dialysis. HSR 2018;53(6):5309-2330.
- 29. The Congressional Budget Office. The health care system for veterans: an interim report. http://www.cbo.gov/ftpdocs/88xx/doc8892/maintext.3.1.shtml. Accessed February 16, 2012.
- 30. Waller D. How VA hospitals became the best. *Time*. 2006;168(10):36-7.
- 31. White R. Former Head of Internal Medicine, Arizona VA. Personal Interview. October 17, 2006.
- 32. Hohnloser SH, Fudim M, Alexander JH, el al. Efficacy and safety of apixaban versus warfarin in patients with atrial fibrillation and extremes in body weight: insights from the ARISTOTLE Trial. *Circulation*. 2019 May 14;139(20):2292-300.
- Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Statist Med. 2015;34:3661-3679.
- Thoemmes F, Ong AD. A primer on inverse probability of treatment weighting and marginal structural models. Curr Epidemiol Rep. 2017;4(1):40-59.
- 35. Leslie S, Thiebaud P. Using propensity scores to adjust for treatment selection bias. SAS Global Forum. 2007.

- Xu S, Ross C, Raebel MA. Use of stabilized inverse propensity scores as weights to directly estimate relative risk and its confidence intervals. *Value Health*. 2010;13(2):273-277.
- 37. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.

#### 14. LIST OF TABLES

| Table 1. | Baseline Demographic and Clinical Characteristic Variables | 17 |
|---|---|---|
| Table 2. | Clinical and Outcome Variables | 20 |
| Table 3. | Power Calculation | 28 |
| Table 4. | Exclusion Criteria | 41 |
| Table 5. | CHADS <sub>2</sub> Score | 44 |
| Table 6. | CHADS2-VASc Score | 47 |
| Table 7. | HAS-BLED Score | 52 |
| Table 8. | Baseline Medication List | 56 |
| Table 9. | Bariatric Surgery Codes | 58 |
| Table 10. | Charlson Comorbidity Index Score Calculation | 63 |
| Table 11. | Baseline Comorbidities | 65 |
| Table 12. | Clinical Outcomes | 69 |
| 15. LIST OF | FIGURES | |
| Figure 1. | Study Design. | 14 |
| 16. ANNEX 1 | . LIST OF STAND ALONE DOCUMENTS | |
| None. | | |

# 17. ANNEX 2. ADDITIONAL INFORMATION

# 17.1. Appendix

Table 4. Exclusion Criteria

| Diagnosis | ICD-9 Code | ICD-10 Code |
|---|---|---|
| Valvular<br>Heart Disease | 394.0, 394.1, 394.2, 394.9, 396.0, 396.1, 396.8, 396.9, 424.0, 745.xx | I050, I051, I052, I058, I059, I080, I088, I089, I340, I341, I342, I348, I349, Q213, Z952, Z953, Z954 |
| Mechanical<br>Heart Valve/<br>Mitral<br>Stenosis<br>(narrow<br>definition) | ICD-9-CM: 996.02, 996.71, 394.0, 394.2, 396.0, 396.1, 746.5 ICD-9 procedure: 35.20, 35.22, 35.24, 36.23, 35.97 CPT: 33405, 92987, 33427, 33426, 33425, 33422, 33420, 33430 | ICD-10 diagnosis codes: T82.01XA, T82.02XA, T82.03XA, T82.09XA, T82.817A- T82.897A, T82.9XXA, I05.0, I05.2, I08.0, Q23.2 ICD-10 Procedure Codes:02RF07Z, 02RF08Z, 02RF0JZ, 02RF0KZ, 02RF37H, 02RF37Z, 02RF38H, 02RF38Z, 02RF3JH, 02RF3JZ, 02RF3KH, 02RF3KZ, 02RF47Z, 02RF48Z, 02RF4JZ, 02RF4KZ, 02RG07Z, 02RG08Z, 02RG0JZ, 02RG0KZ, 02RG37H, 02RG37Z, 02RG38H, 02RG38Z, 02RG3JH, 02RG3JZ, 02RG3KH, 02RG3KZ, 02RG47Z, 02RG48Z, 02RG4JZ, 02RG4KZ, 02RH07Z, 02RG48Z, 02RG4JZ, 02RH0KZ, 02RH07Z, 02RH08Z, 02RH0JZ, 02RH0KZ, 02RH37H, 02RH37Z, 02RH38H, 02RH38Z, 02RH3JH, 02RH3JZ, 02RH3KH, 02RH3KZ, 02RH47Z, 02RH48Z, 02RH4JZ, 02RH4KZ, 02RJ07Z, 02RJ08Z, 02RJ0JZ, 02RJ0KZ, 02RJ47Z, 02RJ48Z, 02RJ4JZ, 02RJ4KZ, 02UG3JZ, X2RF032, X2RF332, X2RF432 |
| VTE | DVT: 451-453, 671.3, 671.4, 671.9; or PE: 415.1, 673.2, 673.8 | I2601, I2602, I2609, I2690, I2692, I2699, I8010, I8011, I8012, I8013, I80201, I80202, I80203, I80209, I80211, I80212, I80213, I80219, I80221, I80222, I80223, I80229, I80231, I80232, I80233, I80239, I80291, I80292, I80293, I80299, I803, I808, I809, I81, I820, I821, I82210, I82211, I82220, I82221, I82290, I82291, I823, I82401, I82402, I82403, I82409, I82411, I82412, I82413, I82419, I82421, I82422, I82423, I82429, I82431, I82432, I82433, I82439, I82441, I82442, I82443, I82449, I82441, I82442, I82443, I82449, I82491, I82492, I82493, I82499, I824Y1, I824Y2, I824Y3, I824Y9, I824Z1, I824Z2, I824Z3, I824Z9, I82501, I82502, I82503, I82509, I82511, I82512, I82513, I82519, I82521, I82522, I82523, I82529, I82531, I82532, I82533, I82539, I82541, I82542, I82543, I82549, I82591, I82592, I82593, I82599, I825Y1, I825Y2, I825Y3, I825Y9, I825Z1, I825Z2, I825Z3, I825Z9, I825Z3, I825Z9, I82601, I82602, I82603, I82609, I82621, I82622, I82623, I82629, I82701, I82702, I82703, I82709, I82711, I82712, I82713, I82719, I82721, I82722, I82723, I82729, I82890, I82891, I8290, I8291, I82821, I82822, I82823, I82829, I82611, I82A22, I82A23, I82A29, I82B11, I82B12, I82B13, I82B19, I82B21, I82B22, I82B23, I82B29, I82C11, I82C12, I82C13, I82C19, I82C21, I82C22, I82C23, I82C29, O871, O88211, O88212, O88213, O88219, O8822, |

| Diagnosis | ICD-9 Code | ICD-10 Code |
|---|---|---|
| | | O8823, T82817A, T82818A |
| Transient AF | Pericarditis: 006.8, 017.9, 036.41, 074.21, 093.81, 098.83, 115.93, 390, 391, 392.0, 393, 411.0, 420.90, 420.91, 420.99, 423.0, 423.1, 423.2, 423.8, 423.9; Hyperthyroidism and Thyrotoxicity: 242.0, 242.1, 242.2, 242.3, 242.4, 242.8, 242.9 | A1884, A3953, A5206, A5483, B3323, E0500, E0501, E0510, E0511, E0520, E0521, E0530, E0531, E0540, E0541, E0580, E0581, E0590, E0591, I010, I011, I012, I018, I019, I020, I092, I241, I300, I301, I308, I309, I310, I311, I312, I313, I318, I319, I32, Z952, Z953, Z954, I300, I301, I308, I309 |
| Valve<br>Replacement<br>Procedure | ICD-9-PCS/HCPCS Codes:<br>35.05-35.09, 35.20-35.28, 35.97 | ICD-10-PCS Codes: 02RF07Z, 02RF08Z, 02RF0JZ, 02RF0KZ, 02RF37H, 02RF37Z, 02RF38H, 02RF38Z, 02RF3JH, 02RF3JZ, 02RF3KH, 02RF3KZ, 02RF47Z, 02RF48Z, 02RF4JZ, 02RF4KZ, 02RG07Z, 02RG08Z, 02RG0JZ, 02RG0KZ, 02RG37H, 02RG37Z, 02RG38H, 02RG38Z, 02RG3JH, 02RG3JZ, 02RG3KH, 02RG3KZ, 02RG47Z, 02RG48Z, 02RG4JZ, 02RG4KZ, 02RH07Z, 02RH08Z, 02RH0JZ, 02RH0KZ, 02RH37H, 02RH37Z, 02RH38H, 02RH38Z, 02RH3JH, 02RH3JZ, 02RH3KH, 02RH3KZ, 02RH47Z, 02RH48Z, 02RH4JZ, 02RH4KZ, 02RJ07Z, 02RJ08Z, 02RJ0JZ, 02RJ0KZ, 02RJ47Z, 02RJ4KZ, 02RJ4ZZ, 02RJ3ZZ, X2RF032, X2RF332, X2RF432 |
| Hip/knee replacement surgery | ICD-9-PCS/HCPCS Codes: 81.40, 81.51, 81.52, 81.53, 81.54, 81.55 | ICD-10-PCS Codes: 0SQ90ZZ, 0SQ93ZZ, 0SQ94ZZ, 0SQ94ZZ, 0SQ9XZZ, 0SQB0ZZ, 0SQB3ZZ, 0SQB4ZZ, 0SQBXZZ, 0SR90J9, 0SR90JA, 0SR90JZ, 0SRB0J9, 0SRB0JA, 0SRB0JZ, 0SRA009, 0SRA00A, 0SRA00Z, 0SRA019, 0SRA01A, 0SRA01Z, 0SRA039, 0SRA03A, 0SRA03Z, 0SRA07Z, 0SRA0J9, 0SRA0JA, 0SRA0JZ, 0SRA07Z, 0SRE009, 0SRE00A, 0SRE00Z, 0SRE019, 0SRE01A, 0SRE01Z, 0SRE039, 0SRE03A, 0SRE03Z, 0SRE07Z, 0SRE0J9, 0SRE0JA, 0SRE0JZ, 0SRE0JZ, 0SRR019, 0SRR01A, 0SRR01Z, 0SRR039, 0SRR03A, 0SRR03Z, 0SRR07Z, 0SRR01A, 0SRR01Z, 0SRR0JZ, 0SRR03Z, 0SRR07Z, 0SRS01Z, 0SRS01Z, 0SRS03A, 0SRS03Z, 0SRS01A, 0SRS01Z, 0SRS01Z, 0SRS0JA, 0SRS0JZ, 0SW93JZ, 0SW94JZ, 0SWB3JZ, 0SWB3JZ, 0SWB4JZ, 0SWB3JZ, 0SWB4JZ, 0SWB3JZ, 0SWB4JZ, 0SWR3JZ, 0SWR3JZ, 0SRS07Z, 0SRS0Z, 0SWB3JZ, 0SWB4JZ, 0SWB3JZ, 0SWB4JZ, 0SWB3JZ, 0SWB4JZ, 0SWB3JZ, 0SWB4JZ, 0SWB3JZ, 0SWB4JZ, 0SRC0Z, 0SRC0Z |

| Diagnosis | ICD-9 Code | ICD-10 Code |
|---|---|---|
| | | 0SWU3JZ, 0SWU4JZ, 0SWV0JZ, 0SWV3JZ, |
| | | 0SWV4JZ, 0SWW0JZ, 0SWW3JZ, 0SWW4JZ |
| Pregnancy | ICD-9 diagnosis codes: 630-679, | ICD- 10 Diagnosis codes: O00-O16, O20-O48, O60- |
| | V22, V23, V24, V27, V28, V61.6, | O77, O80-O82, O85-O92, O94-O9A, Z370, Z371, |
| | V61.7, 792.3, 796.5 | Z372, Z373, Z374, Z3750, Z3751, Z3752, Z3753, |
| | ICD-9 procedure codes: 72.00-75.99 | Z3754, Z3759, Z3760, Z3761, Z3762, Z3763, Z3764, |
| | ICD-9 procedure codes: 72.00-75.99 | Z3769, Z377, Z379, Z36, Z36, Z36, Z36, Z36, Z36, |
| | HCPCS: 59000-59350, 59400-59430, | Z36, Z36, Z36, Z36, Z36, Z640, Z640 |
| | 59510-59866, 59870-59899, 76801- | ICD-10 procedure codes: 102, 109, 10A, 10D, 10E, |
| | 76828, 83661-8366 | 10H. 10J, 10P, 10Q, 10S,10T, 10Y, 2Y44X5Z, |
| | | 30273H1, 30273J1, 30273K1, 30273L1, 30273M1, |
| | | 30273N1, 30273P1, 30273Q1, 30273R1, 30273S1, |
| | | 30273T1, 30273V1, 30273W1, 30277H1, 30277J1, |
| | | 30277K1, 30277L1, 30277M1, 30277N1, 30277P1, |
| | | 30277Q1, 30277R1, 30277S1, 30277T1, 30277V1, |
| | | 30277W1, 3E0DXGC, 3E0E305, 3E0E329, 3E0E33Z, |
| | | 3E0E36Z, 3E0E37Z, 3E0E3BZ, 3E0E3GC, |
| | | 3E0E3HZ, 3E0E3KZ, 3E0E3NZ, 3E0E3SF, |
| | | 3E0E3TZ, 3E0E705, 3E0E729, 3E0E73Z, 3E0E76Z, |
| | | 3E0E77Z, 3E0E7BZ, 3E0E7GC, 3E0E7HZ, |
| | | 3E0E7KZ, 3E0E7NZ, 3E0E7SF, 3E0E7TZ, 3E0E805, |
| | | 3E0E829, 3E0E83Z, 3E0E86Z, 3E0E87Z, 3E0E8BZ, |
| | | 3E0E8GC, 3E0E8HZ, 3E0E8KZ, 3E0E8NZ, |
| | | 3E0E8SF, 3E0E8TZ, 3E0P3VZ, 3E0P7VZ, |
| | | 4A0H74Z, 4A0H7CZ, 4A0H7FZ, 4A0H7HZ, |
| | | 4A0H84Z, 4A0H8CZ, 4A0H8FZ, 4A0H8HZ, |
| | | 4A0HX4Z, 4A0HXCZ, 4A0HXFZ, 4A0HXHZ, |
| | | 4A0J72Z, 4A0J74Z, 4A0J7BZ, 4A0J82Z, 4A0J84Z, |
| | | 4A0J8BZ, 4A0JX2Z, 4A0JX4Z, 4A0JXBZ, |
| | | 4A1H74Z, 4A1H7CZ, 4A1H7FZ, 4A1H7HZ, |
| | | 4A1H84Z, 4A1H8CZ, 4A1H8FZ, 4A1H8HZ, |
| | | 4A1HX4Z, 4A1HXCZ, 4A1HXFZ, 4A1HXHZ, |
| | | 4A1J72Z, 4A1J74Z, 4A1J7BZ, 4A1J82Z, 4A1J84Z, |
| | | 4A1J8BZ, 4A1JX2Z, 4A1JX4Z, 4A1JXBZ |

Table 5. CHADS<sub>2</sub> Score

| CHADS <sub>2</sub> | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| Congestive<br>Heart Failure | 1 | 402.x1, 404.x1, 404.x3,<br>428.xx | I0981, I110, I132, I501, I5020, I5021, I5022, I5023, I5030, I5031, I5032, I5033, I5040, I5041, I5042, I5043, I509 |
| Hypertension | 1 | 401.xx-405.xx | I10, I110, I119, I120, I129, I130, I1310, I1311, I132, I150, I151, I152, I158, I159, I160, I161, I169, N262 |
| Age ≥75 years | 1 | - | - |
| Diabetes mellitus | | 250.xx 357.2, 362.0, 366.41 | E08311, E08319, E083211, E083212, E083213, E083219, E083293, E083299, E083311, E083312, E083313, E083319, E083391, E083392, E083393, E083399, E083411, E083412, E083413, E083419, E083491, E083491, E083492, E083493, E083499, E083511, E083512, E083513, E083519, E083521, E083522, E083523, E083529, E083531, E083529, E083531, E083529, E083531, E083542, E083543, E083549, E083551, E083552, E083553, E083559, E083591, E083552, E083553, E083559, E083591, E083592, E083593, E083599, E0836, E0840, E0842, E09311, E09319, E093211, E093212, E093213, E093293, E093299, E093311, E093312, E093313, E093319, E093391, E093392, E093393, E093399, E093411, E093412, E093413, E093419, E093491, E093491, E093491, E093491, E093512, E093513, E093511, E093512, E093513, E093511, E093512, E093513, E093511, E093512, E093513, E093514, E03314, E103319, E10331411, |

| CHADS <sub>2</sub> | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | | E103412, E103413, E103419, |
| | | | E103491, E103492, E103493, |
| | | | E103499, E103511, E103512, |
| | | | E103513, E103519, E103521, |
| | | | E103522, E103523, E103529, |
| | | | E103531, E103532, E103533, |
| | | | E103539, E103541, E103542, |
| | | | E103543, E103549, E103551, |
| | | | E103552, E103553, E103559, |
| | | | E103591, E103592, E103593, |
| | | | E103599, E1036, E1037X1, E1037X2, |
| | | | E1037X3, E1037X9, E1039, E1040, |
| | | | E1041, E1042, E1043, E1044, E1049, |
| | | | E1051, E1052, E1059, E10610, |
| | | | E10618, E10620, E10621, E10622, |
| | | | E10628, E10630, E10638, E10641, |
| | | | E10649, E1065, E1069, E108, E109, |
| | | | E1100, E1101, E1121, E1122, E1129, |
| | | | E11311, E11319, E113211, E113212, |
| | | | E113213, E113219, E113291, |
| | | | E113292, E113293, E113299, |
| | | | E113311, E113312, E113313, |
| | | | E113319, E113391, E113392, |
| | | | E113393, E113399, E113411, |
| | | | E113412, E113413, E113419, |
| | | | E113491, E113492, E113493,<br>E113499, E113511, E113512, |
| | | | E113513, E113511, E113512,<br>E113513, E113519, E113521, |
| | | | E113513, E113519, E113521,<br>E113522, E113523, E113529, |
| | | | E113522, E113523, E113529,<br>E113531, E113532, E113533, |
| | | | E113531, E113532, E113533,<br>E113539, E113541, E113542, |
| | | | E113543, E113549, E113551, |
| | | | E113552, E113553, E113559, |
| | | | E113591, E113592, E113593, |
| | | | E113599, E1136, E1137X1, E1137X2, |
| | | | E1137X3, E1137X9, E1139, E1140, |
| | | | E1141, E1142, E1143, E1144, E1149, |
| | | | E1151, E1152, E1159, E11610, |
| | | | E11618, E11620, E11621, E11622, |
| | | | E11628, E11630, E11638, E11641, |
| | | | E11649, E1165, E1169, E118, E119, |
| | | | E1300, E1301, E1310, E1311, E1321, |
| | | | E1322, E1329, E13311, E13319, |
| | | | E133211, E133212, E133213, |
| | | | E133219, E133291, E133292, |
| | | | E133293, E133299, E133311, |
| | | | E133312, E133313, E133319, |
| | | | E133391, E133392, E133393, |
| | | | E133399, E133411, E133412, |
| | | | E133413, E133419, E133491, |
| | | | E133492, E133493, E133499, |

| CHADS <sub>2</sub> | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | | E133511, E133512, E133513, E133519, E133521, E133522, E133523, E133529, E133531, E133532, E133533, E133539, E133541, E133542, E133543, E133549, E133551, E133552, E133553, E133559, E133559, E133599, E1336, E1337X1, E1337X2, E1337X3, E1337X1, E1337X2, E1337X3, E1341, E1342, E1343, E1344, E1349, E1351, E1352, E1359, E13610, E13618, E13620, E13621, E13622, E13628, E13630, E13638, E13641, E13649, E1365, E1369, E138, E139, E0851, E0852, E0951, E0952, E1051, E1052, E1151, E1152, E1351, E1352 |
| Stroke | 2 | V12.54, 433-436 | I6300, I63011, I63012, I63013, I63019, I6302, I63031, I63032, I63033, I63039, I6309, I6310, I63111, I63112, I63113, I63119, I6312, I63131, I63132, I63133, I63139, I6319, I6320, I63211, I63212, I63213, I63239, I6329, I63231, I63232, I63233, I63239, I6329, I6330, I63311, I63312, I63313, I63319, I63321, I63322, I63323, I63329, I63331, I63322, I63333, I63339, I63341, I63342, I63343, I63349, I6339, I6340, I63411, I63412, I63423, I63429, I63411, I63422, I63423, I63429, I63431, I63422, I63433, I63439, I6341, I63442, I63443, I63449, I6349, I6350, I63511, I63512, I63513, I63519, I63521, I63522, I63523, I63529, I63531, I63532, I63533, I63539, I63541, I63542, I63543, I63549, I63541, I63542, I63543, I63549, I6359, I6351, I6351, I6502, I6503, I6509, I651, I6521, I6522, I6523, I6529, I658, I659, I6601, I6602, I6603, I6609, I6611, I6612, I6613, I6619, I6621, I6622, I6623, I6629, I663, I668, I669 |

Table 6. CHADS2-VASc Score

| CHA2DS <sub>2</sub> -VASc | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| Congestive Heart<br>Failure | 1 | 402.x1, 404.x1, 404.x3,<br>428.xx | I0981, I110, I132, I501, I5020, I5021, I5022, I5023, I5030, I5031, I5032, I5033, I5040, I5041, I5042, I5043, I509 |
| Hypertension | 1 | 401.xx-405.xx | I10, I110, I119, I120, I129, I130,<br>I1310, I1311, I132, I150, I151, I152,<br>I158, I159, I160, I161, I169, N262 |
| Age ≥75 years | 2 | - | 1-1 |
| Diabetes mellitus | 1 | 250, 357.2, 362.0, 366.41 | E08311, E08319, E083211, E083212, E083213, E083219, E083291, E083292, E083293, E083299, E083311, E083312, E083313, E083319, E083391, E083392, E083393, E083399, E083411, E083412, E083413, E083419, E083491, E083492, E083493, E083499, E083511, E083512, E083513, E083519, E083521, E083522, E083523, E083529, E083531, E083524, E083531, E083532, E083533, E083539, E083541, E083542, E083543, E083544, E083542, E083554, E083552, E083553, E083559, E083591, E083592, E083593, E083599, E083591, E093211, E093212, E093213, E093219, E093291, E093292, E093293, E093299, E093311, E09319, E093291, E093292, E093393, E093399, E093311, E093312, E093392, E093393, E093399, E093411, E093412, E093413, E093414, E093412, E093513, E093592, E093511, E093522, E093531, E093529, E093511, E093522, E093523, E093529, E093531, E093524, E093533, E093529, E093531, E093524, E093542, E093553, E093559, E093593, E093599, E093511, E093512, E093513, E093529, E093511, E093522, E093523, E093529, E093511, E093522, E093523, E093529, E093511, E093522, E093523, E093529, E093511, E093522, E093523, E093529, E093511, E093522, E093523, E093529, E093511, E093522, E093529, E093529, E093529, E093511, E093522, E093529, E033529, E103311, E103312, E1033229, E103313, E103319, E103392, E103392, E103313, E103319, E103392, |

| CHA2DS <sub>2</sub> -VASc | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | | E103393, E103399, E103411, |
| | | | E103412, E103413, E103419, |
| | | | E103491, E103492, E103493, |
| | | | E103499, E103511, E103512, |
| | | | E103513, E103519, E103521, |
| | | | E103522, E103523, E103529, |
| | | | E103531, E103532, E103533, |
| | | | E103539, E103541, E103542, |
| | | | E103543, E103549, E103551, |
| | | | E103552, E103553, E103559, |
| | | | E103591, E103592, E103593, |
| | | | E103599, E1036, E1037X1, |
| | | | E1037X2, E1037X3, E1037X9, |
| | | | E1039, E1040, E1041, E1042, E1043, |
| | | | E1044, E1049, E1051, E1052, E1059, |
| | | | E10610, E10618, E10620, E10621, |
| | | | E10622, E10628, E10630, E10638, |
| | | | E10641, E10649, E1065, E1069, |
| | | | E108, E109, E1100, E1101, E1121, |
| | | | E1122, E1129, E11311, E11319, |
| | | | E113211, E113212, E113213, |
| | | | E113219, E113291, E113292, |
| | | | E113293, E113299, E113311, |
| | | | E113312, E113313, E113319, |
| | | | E113391, E113392, E113393, |
| | | | E113399, E113411, E113412, |
| | | | E113413, E113419, E113491, |
| | | | E113492, E113493, E113499, |
| | | | E113511, E113512, E113513, |
| | | | E113519, E113521, E113522, |
| | | | E113523, E113529, E113531, |
| | | | E113532, E113533, E113539, |
| | | | E113541, E113542, E113543, |
| | | | E113549, E113551, E113552, |
| | | | E113553, E113559, E113591, |
| | | | E113592, E113593, E113599, E1136, |
| | | | E1137X1, E1137X2, E1137X3, |
| | | | E1137X9, E1139, E1140, E1141, |
| | | | E1142, E1143, E1144, E1149, E1151, |
| | | | E1152, E1159, E11610, E11618, |
| | | | E11620, E11621, E11622, E11628, |
| | | | E11630, E11638, E11641, E11649,<br>E1165, E1169, E118, E119, E1300, |
| | | | E1103, E1109, E118, E119, E1300, E1301, E1310, E1311, E1321, E1322, |
| | | | E1301, E1310, E1311, E1321, E1322, E1329, E13311, E13319, E133211, |
| | | | E1329, E13311, E13319, E133211,<br>E133212, E133213, E133219, |
| | | | E133212, E133213, E133219,<br>E133291, E133292, E133293, |
| | | | E133291, E133292, E133293,<br>E133299, E133311, E133312, |
| | | | E133299, E133311, E133312,<br>E133313, E133319, E133391, |
| | | | E133313, E133314, E133391,<br>E133392, E133393, E133399, |
| | | | E133411, E133412, E133413, |
| | | | E133411, E133412, E133413, |

| CHA2DS <sub>2</sub> -VASc | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | | E133419, E133491, E133492,<br>E133493, E133499, E133511,<br>E133512, E133513, E133519,<br>E133521, E133522, E133523,<br>E133529, E133531, E133532,<br>E133533, E133539, E133541,<br>E133542, E133543, E133549,<br>E133551, E133552, E133553,<br>E133559, E133591, E133592,<br>E133593, E133599, E1336, E1337X1,<br>E1337X2, E1337X3, E1337X9,<br>E1339, E1340, E1341, E1342, E1343,<br>E1344, E1349, E1351, E1352, E1359,<br>E13610, E13618, E13620, E13621,<br>E13622, E13628, E13630, E13638,<br>E13641, E13649, E1365, E1369,<br>E138, E139, E0851, E0852, E0951,<br>E0952, E1051, E1052, E1151, E1152,<br>E1351, E1352 |
| Stroke (non-hemorrhagic only & transient ischemic attack) | 2 | V12.54, 433.xx-436.xx | I6300, I63011, I63012, I63013, I63019, I6302, I63031, I63032, I63033, I63039, I6309, I6310, I63111, I63112, I63113, I63131, I63131, I63132, I63133, I63139, I6319, I6320, I63211, I63212, I63213, I63219, I6322, I63231, I63232, I63233, I63239, I6329, I6330, I63311, I63312, I63313, I63319, I63321, I63322, I63323, I63329, I63321, I63322, I63333, I63339, I63331, I63332, I63333, I63339, I63341, I63342, I63343, I63349, I63341, I63412, I63413, I63419, I63421, I63422, I63423, I63429, I63431, I63442, I63443, I63449, I63441, I63442, I63443, I63449, I6349, I6350, I63511, I63512, I63513, I63519, I63521, I63522, I63523, I63529, I63531, I63542, I63543, I63549, I63541, I63542, I63543, I63549, I6359, I636, I638, I639, I6501, I6502, I6503, I6509, I651, I6521, I6522, I6523, I6529, I658, I659, I6601, I6602, I6603, I6609, I6611, I6612, I6613, I6619, I6621, I6622, I6623, I6629, I663, I668, I669 |
| Vascular Disease<br>(myocardial<br>infarction,<br>peripheral arterial<br>disease, aortic | 1 | 410.xx, 412, 440.xx, 441.xx,<br>442.xx, 443.xx, 444.2x,<br>445.0x | I200, I2101, I2102, I2109, I2111, I2119, I2121, I2129, I213, I214, I220, I221, I222, I228, I229, I240, I241, I248, I249, I25110, I252, I25700, I25710, I25720, I25730, I25750, |

| CHA2DS <sub>2</sub> -VASc | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| plaque) | | | I25760, I25790, I670, I700, I701, |
| 13050 13500 Selice | | | I70201, I70202, I70203, I70208, |
| | | | 170209, 170211, 170212, 170213, |
| | | | I70218, I70219, I70221, I70222, |
| | | | 170223, 170228, 170229, 170231, |
| | | | 170232, 170233, 170234, 170235, |
| | | | 170238, 170239, 170241, 170242, |
| | | | 170243, 170244, 170245, 170248, |
| | | | 170249, 17025, 170261, 170262, |
| | | | 170263, 170268, 170269, 170291, |
| | | | 170292, 170293, 170298, 170299, |
| | | | 170301, 170302, 170303, 170308, |
| | | | 170309, 170311, 170312, 170313, |
| | | | 170318, 170319, 170321, 170322, |
| | | | 170323, 170328, 170329, 170331, |
| | | | 170332, 170333, 170334, 170335, |
| | | | 170338, 170339, 170341, 170342, |
| | | | 170343, 170344, 170345, 170348, |
| | | | 170349, 17035, 170361, 170362, |
| | | | 170363, 170368, 170369, 170391, |
| | | | 170392, 170393, 170398, 170399, |
| | | | 170401, 170402, 170403, 170408, |
| | | | 170409, 170411, 170412, 170413, |
| | | | 170418, 170419, 170421, 170422, |
| | | | 170423, 170428, 170429, 170431, |
| | | | 170432, 170433, 170434, 170435, |
| | | | 170438, 170439, 170441, 170442, |
| | | | 170443, 170444, 170445, 170448, |
| | | | 170449, 17045, 170461, 170462, |
| | | | 170463, 170468, 170469, 170491, |
| | | | 170492, 170493, 170498, 170499, |
| | | | 170501, 170502, 170503, 170508, |
| | | | 170509, 170511, 170512, 170513, |
| | | | 170518, 170519, 170521, 170522, |
| | | | 170523, 170528, 170529, 170531, |
| | | | 170532, 170533, 170534, 170535, |
| | | | 170538, 170539, 170541, 170542, |
| | | | 170543, 170544, 170545, 170548, |
| | | | 170549, 17055, 170561, 170562, |
| | | | 170563, 170568, 170569, 170591, |
| | | | 170592, 170593, 170598, 170599, |
| | | | 170601, 170602, 170603, 170608, |
| | | | I70609, I70611, I70612, I70613, |
| | | | 170618, 170619, 170621, 170622, |
| | | | 170623, 170628, 170629, 170631, |
| | | | 170632, 170633, 170634, 170635, |
| | | | 170638, 170639, 170641, 170642, |
| | | | 170643, 170644, 170645, 170648, |
| | | | 170649, 17065, 170661, 170662, |
| | | | 170663, 170668, 170669, 170691, |
| | | | 170692, 170693, 170698, 170699, |

| CHA2DS <sub>2</sub> -VASc | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | | 170701, 170702, 170703, 170708, |
| | | | 170709, 170711, 170712, 170713, |
| | | | 170718, 170719, 170721, 170722, |
| | | | 170723, 170728, 170729, 170731, |
| | | | 170732, 170733, 170734, 170735, |
| | | | 170738, 170739, 170741, 170742, |
| | | | 170743, 170744, 170745, 170748, |
| | | | 170749, 17075, 170761, 170762, |
| | | | 170763, 170768, 170769, 170791, |
| | | | 170792, 170793, 170798, 170799, 1708, |
| | | | 17090, 17091, 17092, 17100, 17101, |
| | | | 17102, 17103, 1711, 1712, 1713, 1714, |
| | | | 1715, 1716, 1718, 1719, 1720, 1721, |
| | | | 1722, 1723, 1724, 1725, 1726, 1728, |
| | | | 1729, 17300, 17301, 1731, 17381, |
| | | | 17389, 1739, 1742, 1743, 1744, 175011, |
| | | | 175012, 175013, 175019, 175021, |
| | | | 175022, 175023, 175029, 17770, 17771, |
| | | | 17772, 17773, 17774, 17775, 17776, |
| | | | 17777, 17779, 1790, 1791, 1798 |
| Age | 1 | Age 65-75 years | y <del>-</del> 1 |
| Sex Category | 1 (Female) | 2 | - |

Table 7. HAS-BLED Score

| HAS-BLED | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| Hypertension | 1 point | 401.xx-405.xx | I10, I110, I119, I120, I129, I130, I1310, I1311, I132, I150, I151, I152, I158, I159, I160, I161, I169, N262 |
| Abnormal kidney and/or liver function: | 1 point each | Kidney: 580.xx-589.xx | B520, E0821, E0822, E0829, E0921, E0922, E0929, M3214, M3215, M3504, N000, N001, N002, N003, N004, N005, N006, N007, N008, N009, N010, N011, N012, N013, N014, N015, N016, N017, N018, N019, N020, N021, N022, N023, N024, N025, N026, N027, N030, N031, N032, N033, N034, N035, N036, N037, N038, N039, N040, N041, N042, N043, N044, N045, N046, N047, N048, N049, N050, N051, N052, N053, N054, N055, N056, N057, N058, N059, N060, N061, N062, N063, N064, N065, N060, N061, N062, N063, N064, N065, N066, N067, N068, N069, N070, N071, N072, N073, N074, N075, N076, N077, N078, N079, N08, N140, N141, N142, N143, N144, N150, N158, N159, N16, N170, N171, N172, N178, N179, N181, N182, N183, N184, N185, N186, N189, N19, N250, N251, N2581, N2589, N259, N261, N269, N270, N271, N279 |
| Age ≥75 years | 2 | Liver: 570.xx-573.xx | B251, K700, K7010, K7011, K702, K7030, K7031, K7040, K7041, K709, K710, K7110, K7111, K712, K713, K714, K7150, K7151, K716, K717, K718, K719, K7200, K7201, K7210, K7211, K7290, K7291, K730, K731, K732, K738, K739, K740, K741, K742, K743, K744, K745, K7460, K7469, K750, K751, K752, K753, K754, K7581, K7589, K759, K760, K761, K762, K763, K764, K765, K766, K767, K7681, K7689, K769, K77 |
| Stroke | 1 point | History of stroke V12.54,<br>433.xx-436.xx | G450, G451, G452, G458, G459,<br>G460, G461, G462, I6300, I63011,<br>I63012, I63013, I63019, I6302,<br>I63031, I63032, I63033, I63039,<br>I6309, I6310, I63111, I63112, |

| HAS-BLED | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | | I63113, I63119, I6312, I63131, I63132, I63133, I63139, I6319, I6320, I63211, I63212, I63213, I63219, I6322, I63231, I63232, I63233, I63239, I6329, I6330, I63311, I63312, I63323, I63329, I63321, I63322, I63323, I63329, I63331, I63332, I63333, I63339, I63341, I63342, I63343, I63349, I63341, I63342, I63441, I63412, I63413, I63419, I63421, I63422, I63423, I63429, I63431, I63432, I63433, I63439, I63441, I63442, I63443, I63449, I6349, I6350, I63511, I63512, I63513, I63519, I63521, I63522, I63523, I63529, I63531, I63542, I63543, I63549, I6359, I636, I638, I639, I6501, I6502, I6503, I6509, I651, I6521, I6522, I6523, I6659, I6601, I6602, I6603, I6609, I6611, I6612, I6613, I6619, I6621, I6622, I6623, I6629, I663, I668, I669, I67841, I67848, Z8673 |
| Bleeding | 1 point | Baseline bleeding (Table 12) and 280.xx-286.xx | A985, D500, D508, D509, D510, D511, D512, D513, D518, D519, D520, D521, D528, D529, D530, D531, D552, D553, D558, D559, D550, D551, D552, D553, D558, D559, D560, D561, D562, D563, D565, D568, D569, D5700, D5701, D5702, D571, D5720, D57211, D57212, D57219, D573, D5740, D57411, D57412, D57419, D5780, D57811, D57812, D57819, D580, D581, D582, D588, D589, D590, D591, D592, D593, D594, D595, D596, D598, D599, D600, D601, D608, D609, D6101, D6109, D611, D612, D613, D61810, D61811, D61818, D6182, D649, D65, D66, D67, D680, D681, D682, D684, D649, D65, D66, D67, D680, D681, D682, D68311, D68312, D68318, D6832, D684, D688, D689, D7801, D7802, D7821, D7822, E3601, E3602, E89810, E89811, G9731, G9732, |

| G9751, G9752, H0<br>H05233, H05239,<br>H1132, H1133, H2<br>H2102, H2103, H3<br>H31303, H31309, | H1130, H1131, |
|---|---|
| H1132, H1133, H2<br>H2102, H2103, H3 | |
| H2102, H2103, H3 | 2100, H2101, |
| H31303 H31309 | 31301, H31302, |
| H31312, H31313, | |
| H31411, H31412, | H31413, |
| H31419, H3560, H | |
| H3563, H35731, H | |
| H35733, H35739, | |
| H4312, H4313, H4 | |
| H44813, H44819, | |
| H47022, H47023, | 1010 G (1) C (1) C (1) |
| H59111, H59112, | |
| H59119, H59121, | |
| H59123, H59129, | |
| H59312, H59313, | 5 |
| H59321, H59322, | 5) |
| H59329, H61121, | |
| H61123, H61129, | |
| H9541, H9542, I31 | |
| I6001, I6002, I601 | |
| 1602, 16030, 16031 | |
| I6050, I6051, I605 | |
| I608, I609, I610, Id | |
| I614, I615, I616, Id | |
| I6200, I6201, I620 | |
| I629, I8501, I8511 | |
| I97411, I97418, I9 | |
| 197611, 197618, 19 | |
| J9562, J95830, J95 | 하다 하는 사람들이 들었다. 안 살아 하다 살폈다. |
| K226, K250, K252<br>K260, K262, K264 | 15 (5) |
| K200, K202, K204<br>K272, K274, K276 | |
| K272, K274, K276<br>K284, K286, K290 | 70 O O |
| K294, K290, K290<br>K2931, K2941, K2 | |
| K2931, K2941, K2<br>K2971, K2981, K2 | |
| K3182, K5521, K5 | |
| K5162, K3521, K5<br>K5713, K5721, K5 | |
| K5741, K5751, K5 | |
| K5791, K5793, K6 | |
| K640, K641, K642 | 50 50 |
| K661, K9161, K91 | |
| K91841, K920, K9 | |
| L7601, L7602, L76 | |
| M2500, M25011, I | |
| M25019, M25021, | |
| M25029, M25031, | |
| M25039, M25041, | |
| M25049, M25051, | |
| M25059, M25061, | |

| HAS-BLED | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| HAS-BLED | Point | ICD-9 Codes | M25069, M25071, M25072, M25073, M25074, M25075, M25076, M2508, M96810, M96811, M96830, M96831, N421, N837, N857, N920, N9961, N9962, N99820, N99821, R040, R041, R042, R0489, R049, R310, R319, R58, R710, S0190XA, S062X0A, S062X1A, S062X2A, S062X3A, S062X4A, S062X5A, S062X6A, S062X7A, S062X8A, S062X9A, S06300A, S06301A, S06302A, S06303A, S06304A, S06305A, S06306A, S06307A, S06308A, S06309A, S06340A, S06341A, S06342A, S06343A, S06347A, S06348A, S06349A, S06350A, S06351A, S06352A, S06350A, S06351A, S06355A, S06356A, S06357A, S06358A, S063636A, S0636A, S06361A, S0636A, S0636A, S0636A, S0635A, S0635A, S0636A, S0635A, S0636A, S0635A, S0635A, S0636A, S0635A, S0636A, S0636A, S0635A, S0636A, S0636A, S0635A, S0635A, S0636A, S0635A, S0635A, S0636A, S0635A, S0636A, S0636A, S0635A, S0636A, S0636A, S0635A, S0636A, S0636A, S0635A, S0635A, S0636AA, S0635A, S0636A, S0636AA, S0635A, S0636A, S0636AA, S0635A, S0636A, S0636AA, S0635A, S0635AA, S0636AA, S0635A, S0636AA, S0636AA, S0635A, S0636AA, S0636AA, S0635A, S0636AA, S064X0A, S064XAA, S064XSA, S064XAA, S064XAA, S064XSA, S064XAA, S065XAA, S066XAA, S066XSA, S066XAA, S066XAA, S066XSA, S068YA, S068YAA, S069XAA, S069XAA, S069XSA, S069XAA, |
| | | | S069X9A, S36112A, S37021A,<br>S37022A, S37029A, T792XXA |
| Labile INR | Not applicable | Not measurable. | Not applicable |
| Elderly | 1 point for<br>age 65 or older | 65+ years | 65+ years |
| Alcohol/ Drug<br>Therapy | 1 point | 303.xx, 305.0x, V11.3x<br><u>Antiplatelets administered</u><br>(abciximab, anagrelide HCL,<br>aspirin, aspirin/dipyridamole, | F1010, F10120, F10129, F1020,<br>F1021, F10220, F10229 |

| HAS-BLED | Point | ICD-9 Codes | ICD-10 Codes |
|---|---|---|---|
| | | cilostazol, clopidogrel, dipyridamole, eptifibatide, prasugrel, ticagrelor, ticlopidine, tirofiban) NSAIDs administered (bromfenac, celecoxib, diclofenac, etodolac, fenoprofen, flurbiprofen, ibuprofen, indomethacin, ketoprofen, ketorolac, lansoprazole/naproxen, meclofenamate, mefenamic acid, meloxicam, nabumetone, naproxen, oxaprozin, piroxicam, sulindac, tolmetin) | |

### Table 8. Baseline Medication List

| Mechanism of<br>Action | | Drug |
|---|---|---|
| Angiotensin<br>converting enzyme<br>inhibitor | Benazepril, Captopril, Enalapril, Fosinopril, Lisinopril, Moexipril, Perindopril, Quinapril, Ramipril, Trandolapril | |
| Amiodarone | Amiodarone | |
| Angiotensin receptor blocker | Azilsartan, Can<br>Valsartan | desartan, Eprosartan, Irbesartan, Losartan, Olmesartan, Telmisartan, |
| Beta blockers | Acebutolol, Atenolol, Betaxolol, Bisoprolol, Esmolol, Carteolol, Carvedeolol, Labetalol, Levobunolol, Metipranolol, Metoprolol, Nebivolol, Nadolol, Penbutolol, Pinodolol, Propranolol, Sotalal, Timolol, | |
| H2-receptor antagonist | Burimamide, Cimetidine, Ebrotidine, Famotidine, Metiamide, Nizatidine, Ranitidine | |
| Proton pump inhibitor | Lansoprazole, Omeprazole, Pantoprazole, Rabeprazole, Dexlansoprazole, Esomeprazole | |
| Statins | Atorvastatin, Fluvastatin, Lovastatin, Pitavastatin, Pravastatin, Rosuvastatin, Simvastatin. | |
| Anti-platelets | Aspirin, Clopidogrel, Prasugrel, Ticlopidine, Cilostazol, Abciximab, Epifibatide, Tirofiban, Dipyridamole, Ticagrelor | |
| Inhibitors of Warfarin | CYP2C9<br>inhibitors | amiodarone, capecitabine, cotrimoxazole, etravirine, fluconazole, fluvastatin, fluvoxamine, metronidazole, miconazole, oxandrolone, sulfinpyrazone, tigecycline, voriconazole, zafirlukast |
| | CYP1A2 inhibitors | acyclovir, allopurinol, caffeine, cimetidine, ciprofloxacin, disulfiram, enoxacin, famotidine, fluvoxamine, methoxsalen, mexiletine, norfloxacin, oral contraceptives (ethinyl estradiol, levonorgestrel, desogestrel, norethindrone, norgestrel, mestranol, |

| Mechanism of<br>Action | Drug | |
|---|---|---|
| | | drospirenone), phenylpropanolamine, propafenone, propranolol, terbinafine, thiabendazole, ticlopidine, verapamil, zileuton |
| | CYP3A4 inhibitors | alprazolam, amiodarone, amlodipine, amprenavir, aprepitant, atorvastatin, atazanavir, bicalutamide, cilostazol, cimetidine, ciprofloxacin, clarithromycin, conivaptan, cyclosporine, darunavir/ritonavir, diltiazem, erythromycin, fluconazole, fluoxetine, fluvoxamine, fosamprenavir, imatinib, indinavir, isoniazid, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, nilotinib, oral contraceptives (ethinyl estradiol, levonorgestrel, desogestrel, norethindrone, norgestrel, mestranol, drospirenone), posaconazole, ranitidine, ranolazine, ritonavir, saquinavir, telithromycin, tipranavir, voriconazole, zileuton |
| Inducers of Warfarin | CYP2C9<br>inducers | aprepitant, bosentan, carbamazepine, phenobarbital, rifampin |
| | CYP1A2<br>inducers | montelukast, moricizine, omeprazole, phenobarbital, phenytoin |
| | CYP3A4 inducers | armodafinil, amprenavir, aprepitant, bosentan,<br>carbamazepine, efavirenz, etravirine, modafinil, nafcillin,<br>phenytoin, prednisone, rifampin, rufinamide |
| Dronedarone | dronedarone | |
| Digoxin | digoxin; J1160; J1162 | |
| Calcium Channel<br>Blockers | diltiazem, felodipine, Isradipine, nicardipine, nisoldipine, verapamil, amlodipine, bepridil, clevidipine, mibefradil, nifedipine and nimodipine | |
| Renin Angiotensin<br>System Antagonists | benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan, azilsartan, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan, eplerenone, spironolactone | |
| Glucocorticoids [oral and injectable] | beclomethasone, betamethasone, budesonide, cortisone, dexamethasone, hydrocortisone, methylprednisolone, prednisolone, prednisone, triamcinolone | |
| Diuretics | acetazolamide, methazolamide, bumetanide, ethacrynic acid, torsemide, furosemide, pamabrom, eplerenone, triamterene, spironolactone, amiloride, indapamide, hydrochlorothiazide, chlorthalidone, metolazone, methyclothiazide, bendroflumethiazide, polythiazide | |
| Metformin | Metformin | |
| Sulfonylureas | acetohexamide, chlorpropamide, glimepiride, glipizide, glyburide, tolazamide, tolbutamide | |
| Thiazolidinedione | pioglitazone, rosiglitazone | |
| Insulin | insulin | |

| Mechanism of<br>Action | Drug |
|---|---|
| Other Diabetes Drugs | exenatide, liraglutide, dulaglutide, repaglinide, sitagliptin, saxagliptin, linagliptin, alogliptin, nateglinide, acarbose, miglitol, canagliflozin, dapagliflozin, empagliflozin, pramlintide |
| Antiulcer Agents | nitzatidine, sucralfate, misoprostol, famotidine, omeprazole, cimetidine, ranitidine hydrochloride, Dexlansoprazole, Esomeprazole, Lansoprazole, Omeprazole, Pantoprazole, Rabeprazole, Burimamide, Ebrotidine, Metiamide, Cisapride, Pirenzepine, Propantheline, Roxatidine acetate |
| Antidepressant | citalopram, escitalopram, paroxetine, fluoxetine, fluvoxamine, sertraline, desvenlafaxine, duloxetine, levomilnacipran, milnacipran, venlafaxine, vilazodone, vortioxetine, nefazodone, trazodone, reboxetine, teniloxazine, viloxazine, bupropion, amitriptyline, amitriptylinoxide, clomipramine, desipramine, dibenzepin, dimetacrine, dosulepin, doxepin, imipramine, lofepramine, melitracen, nitroxazepine, nortriptyline, noxiptiline, opipramol, pipofezine, protriptyline, trimipramine, amoxapine, maprotiline, mianserin, mirtazapine, setiptiline, isocarboxazid, phenelzine, tranylcypromine, selegiline, caroxazone, metralindole, moclobemide, pirlindole, toloxatone, bifemelane, amisulpride, lurasidone, quetiapine, aripiprazole, brexpiprazole, lurasidone, olanzapine, quetiapine, risperidone, lithium |

Table 9. Bariatric Surgery Codes

| Туре | Codes | Description |
|---|---|---|
| СРТ | 43842 | Gastric restrictive procedure without gastric bypass for morbid obesity; vertical-banded gastroplasty |
| | 43843 | Gastric restrictive procedure without gastric bypass for morbid obesity; other than vertical-banded gastroplasty |
| | 43846 | Gastric restrictive procedure with gastric bypass for morbid obesity with short limb Roux-en-y gastroenterostomy |
| | 43847 | Gastric restrictive procedure with gastric bypass for morbid obesity with small intestine reconstruction to limit absorption |
| | 43848 | Revision of gastric restrictive procedure for morbid obesity |
| | 43659 | Unlisted laparoscopic procedure, stomach |
| | 43644 | Laparoscopy, surgical, gastric restrictive procedure; with gastric bypass and Roux-en-Y gastroenterostomy |
| | 43844 | Laparoscopic gastric restrictive procedure with gastric bypass and<br>Roux- en-Y gastroenterostomy |
| | S2085 | laparoscopic gastric bypass |
| | 43645 | Laparoscopy, surgical, gastric restrictive procedure; with gastric bypass and small intestine reconstruction to limit absorption |
| | 43770 | Laparoscopy, surgical, gastric restrictive procedure; placement of adjustable gastric band |

| Type | Codes | Description |
|---|---|---|
| | 43771 | Revision of adjustable gastric band component only |
| | 43773 | Laparoscopy, surgical, gastric restrictive procedure; removal and replacement of adjustable gastric restrictive device component only |
| | S2082 | Laparoscopy, surgical; gastric restrictive procedure, adjustable gastric band includes placement of subcutaneous port |
| ICD-9 diagnosis | V45.86 | Bariatric surgery status |
| ICD-10 diagnosis | Z98.84 | Bariatric surgery status |
| ICD-9 procedure | 43.89 | Open and other partial gastrectomy |
| | 44.31 | High gastric bypass |
| | 44.38 | Laparoscopic gastroenterostomy |
| | 44.39 | Other gastroenterostomy without gastrectomy |
| | 44.68 | Laparoscopic gastroplasty |
| | 44.95 | Laparoscopic gastric restrictive procedure |
| | 44.96 | Laparoscopic Revision of Gastric Restrictive Procedure |
| | 44.97 | Laparoscopic Removal of Gastric Restrictive Device(s) |
| | 44.99 | Other Operations on Stomach |
| | 44.5 | Revision of Gastric Anastomosis |
| | 45.51 | Isolation of Segment of Small Intestine |
| | 45.9 | Intestinal Anastomosis |
| ICD-10 procedure | 0D16079 | Bypass Stomach to Duodenum with Autologous Tissue Substitute,<br>Open Approach |
| | 0D1607A | Bypass Stomach to Jejunum with Autologous Tissue Substitute, Open<br>Approach |
| | 0D160J9 | Bypass Stomach to Duodenum with Synthetic Substitute, Open<br>Approach |
| | 0D160JA | Bypass Stomach to Jejunum with Synthetic Substitute, Open Approach |
| | 0D160K9 | Bypass Stomach to Duodenum with Nonautologous Tissue Substitute,<br>Open Approach |
| | 0D160KA | Bypass Stomach to Jejunum with Nonautologous Tissue Substitute,<br>Open Approach |
| | 0D160Z9 | Bypass Stomach to Duodenum, Open Approach |
| | 0D160ZA | Bypass Stomach to Jejunum, Open Approach |
| | 0D160ZB | Bypass Stomach to Ileum, Open Approach |
| | 0D16479 | Bypass Stomach to Duodenum with Autologous Tissue Substitute,<br>Percutaneous Endoscopic Approach |
| | 0D1647A | Bypass Stomach to Jejunum with Autologous Tissue Substitute, |

| Type | Codes | Description |
|---|---|---|
| | | Percutaneous Endoscopic Approach |
| | 0D164J9 | Bypass Stomach to Duodenum with Synthetic Substitute, Percutaneous<br>Endoscopic Approach |
| | 0D164JA | Bypass Stomach to Jejunum with Synthetic Substitute, Percutaneous<br>Endoscopic Approach |
| | 0D164K9 | Bypass Stomach to Duodenum with Nonautologous Tissue Substitute,<br>Percutaneous Endoscopic Approach |
| | 0D164KA | Bypass Stomach to Jejunum with Nonautologous Tissue Substitute,<br>Percutaneous Endoscopic Approach |
| | 0D164Z9 | Bypass Stomach to Duodenum, Percutaneous Endoscopic Approach |
| | 0D164ZA | Bypass Stomach to Jejunum, Percutaneous Endoscopic Approach |
| | 0D16879 | Bypass Stomach to Duodenum with Autologous Tissue Substitute, Via<br>Natural or Artificial Opening Endoscopic |
| | 0D1687A | Bypass Stomach to Jejunum with Autologous Tissue Substitute, Via<br>Natural or Artificial Opening Endoscopic |
| | 0D168J9 | Bypass Stomach to Duodenum with Synthetic Substitute, Via Natural or Artificial Opening Endoscopic |
| | 0D168JA | Bypass Stomach to Jejunum with Synthetic Substitute, Via Natural or<br>Artificial Opening Endoscopic |
| | 0D168K9 | Bypass Stomach to Duodenum with Nonautologous Tissue Substitute,<br>Via Natural or Artificial Opening Endoscopic |
| | 0D168KA | Bypass Stomach to Jejunum with Nonautologous Tissue Substitute,<br>Via Natural or Artificial Opening Endoscopic |
| | 0D168Z9 | Bypass Stomach to Duodenum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D168ZA | Bypass Stomach to Jejunum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0DB60ZZ | Excision of Stomach, Open Approach |
| | 0DB63ZZ | Excision of Stomach, Percutaneous Approach |
| | 0DB67ZZ | Excision of Stomach, Via Natural or Artificial Opening |
| | 0DB80ZZ | Excision of Small Intestine, Open Approach |
| | 0DB90ZZ | Excision of Duodenum, Open Approach |
| | 0DBB0ZZ | Excision of Ileum, Open Approach |
| | 0DP643Z | Removal of Infusion Device from Stomach, Percutaneous Endoscopic<br>Approach |
| | 0DP64CZ | Removal of Extraluminal Device from Stomach, Percutaneous<br>Endoscopic Approach |
| | 0DQ60ZZ | Repair Stomach, Open Approach |

| Type | Codes | Description |
|---|---|---|
| | 0DQ63ZZ | Repair Stomach, Percutaneous Approach |
| | 0DQ64ZZ | Repair Stomach, Percutaneous Endoscopic Approach |
| | 0DQ67ZZ | Repair Stomach, Via Natural or Artificial Opening |
| | 0DQ68ZZ | Repair Stomach, Via Natural or Artificial Opening Endoscopic |
| | 0DV64CZ | Restriction of Stomach with Extraluminal Device, Percutaneous<br>Endoscopic Approach |
| | 0DW643Z | Revision of Infusion Device in Stomach, Percutaneous Endoscopic<br>Approach |
| | 0DW64CZ | Revision of Extraluminal Device in Stomach, Percutaneous<br>Endoscopic Approach |
| | 0D190Z9 | Bypass Duodenum to Duodenum, Open Approach |
| | 0D190ZA | Bypass Duodenum to Jejunum, Open Approach |
| | 0D190ZB | Bypass Duodenum to Ileum, Open Approach |
| | 0D190ZL | Bypass Duodenum to Transverse Colon, Open Approach |
| | 0D194Z9 | Bypass Duodenum to Duodenum, Percutaneous Endoscopic Approach |
| | 0D194ZA | Bypass Duodenum to Jejunum, Percutaneous Endoscopic Approach |
| | 0D194ZB | Bypass Duodenum to Ileum, Percutaneous Endoscopic Approach |
| | 0D194ZL | Bypass Duodenum to Transverse Colon, Percutaneous Endoscopic<br>Approach |
| | 0D198Z9 | Bypass Duodenum to Duodenum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D198ZA | Bypass Duodenum to Jejunum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D198ZB | Bypass Duodenum to Ileum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D198ZL | Bypass Duodenum to Transverse Colon, Via Natural or Artificial<br>Opening Endoscopic |
| | 0D1A0ZA | Bypass Jejunum to Jejunum, Open Approach |
| | 0D1A0ZB | Bypass Jejunum to Ileum, Open Approach |
| | 0D1A0ZH | Bypass Jejunum to Cecum, Open Approach |
| | 0D1A0ZK | Bypass Jejunum to Ascending Colon, Open Approach |
| | 0D1A0ZL | Bypass Jejunum to Transverse Colon, Open Approach |
| | 0D1A0ZM | Bypass Jejunum to Descending Colon, Open Approach |
| | 0D1A0ZN | Bypass Jejunum to Sigmoid Colon, Open Approach |
| | 0D1A0ZP | Bypass Jejunum to Rectum, Open Approach |
| | 0D1A4ZA | Bypass Jejunum to Jejunum, Percutaneous Endoscopic Approach |

| Type | Codes | Description |
|---|---|---|
| | 0D1A4ZB | Bypass Jejunum to Ileum, Per cutaneous Endoscopic Approach |
| | 0D1A4ZH | Bypass Jejunum to Cecum, Per cutaneous Endoscopic Approach |
| | 0D1A4ZK | Bypass Jejunum to Ascending Colon, Percutaneous Endoscopic<br>Approach |
| | 0D1A4ZL | Bypass Jejunum to Transverse Colon, Percutaneous Endoscopic<br>Approach |
| | 0D1A4ZM | Bypass Jejunum to Descending Colon, Percutaneous Endoscopic<br>Approach |
| | 0D1A4ZN | Bypass Jejunum to Sigmoid Colon, Percutaneous Endoscopic<br>Approach |
| | 0D1A4ZP | Bypass Jejunum to Rectum, Percutaneous Endoscopic Approach |
| | 0D1A8ZA | Bypass Jejunum to Jejunum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1A8ZB | Bypass Jejunum to Ileum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1A8ZH | Bypass Jejunum to Cecum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1A8ZK | Bypass Jejunum to Ascending Colon, Via Natural or Artificial Opening Endoscopic |
| | 0D1A8ZL | Bypass Jejunum to Transverse Colon, Via Natural or Artificial<br>Opening Endoscopic |
| | 0D1A8ZM | Bypass Jejunum to Descending Colon, Via Natural or Artificial<br>Opening Endoscopic |
| | 0D1A8ZN | Bypass Jejunum to Sigmoid Colon, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1A8ZP | Bypass Jejunum to Rectum, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1B0ZB | Bypass Ileum to Ileum, Open Approach |
| | 0D1B0ZH | Bypass Ileum to Cecum, Open Approach |
| | 0D1B0ZK | Bypass Ileum to Ascending Colon, Open Approach |
| | 0D1B0ZL | Bypass Ileum to Transvers e Colon, Open Approach |
| | 0D1B0ZM | Bypass Ileum to Descending Colon, Open Approach |
| | 0D1B4ZN | Bypass Ileum to Sigmoid Colon, Percutaneous Endoscopic Approach |
| | 0D1B4ZP | Bypass Ileum to Rectum, Percutaneous Endoscopic Approach |
| | 0D1B4ZQ | Bypass Ileum to Anus, Percutaneous Endoscopic Approach |
| | 0D1B8ZB | Bypass Ileum to Ileum, Via Natural or Artificial Opening Endoscopic |
| | 0D1B8ZH | Bypass Ileum to Cecum, Vi a Natural or Artificial Opening Endoscopic |

| Type | Codes | Description |
|---|---|---|
| | 0D1B8ZK | Bypass Ileum to Ascending Colon, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1B8ZL | Bypass Ileum to Transvers e Colon, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1B8ZM | Bypass Ileum to Descending Colon, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1B8ZN | Bypass Ileum to Sigmoid Colon, Via Natural or Artificial Opening<br>Endoscopic |
| | 0D1B8ZP | Bypass Ileum to Rectum, Via Natural or Artificial Opening Endoscopic |
| | 0D1B8ZQ | Bypass Ileum to Anus, Via Natural or Artificial Opening Endoscopic |

Table 10. Charlson Comorbidity Index Score Calculation

| Condition | ICD-9 Code(s) | ICD-10 Code(s) | Point |
|---|---|---|---|
| Myocardial<br>Infarction | 410.xx; 412.xx | I21, I22, I252 | 1 |
| Congestive Heart<br>Failure | 428.xx | I43, I50, I099, I110, I130, I132, I255, I420, I425, I426, I427, I428, I429, P290 | 1 |
| Peripheral<br>vascular disease | 441.xx; 443.9x; 785.4x; v43.4x,<br>procedure: 38.48 | I70, I71, I731, I738, I739, I771, I790, I792, K551, K558, K559, Z958, Z959 | 1 |
| Cerebrovascular<br>disease | 430.xx-438.99<br>Modified to remove 430.xx-432.xx | G45, G46, I60, I61, I62, I63, I64, I65, I66, I67, I68, I69, H340 | 1 |
| Dementia | 290.xx | F00, F01, F02, F03, G30, F051, G311 | 1 |
| Chronic<br>obstructive<br>pulmonary<br>disease | 490.xx-496.99; 500.xx-505.99;<br>506.4x | J40, J41, J42, J43, J44, J45, J46, J47, J60, J61, J62, J63, J64, J65, J66, J67, I278, I279, J684, J701, J703 | 1 |
| Rheumatologic<br>disease | 710.0x-710.19; 710.4x-; 714.0x-<br>714.29; 714.81; 725.xx | M05, M32, M33, M34, M06, M315,<br>M351, M353, M360 | 1 |
| Peptic ulcer<br>disease | 531.0x-531.79; 532.4x-532.79;<br>533.4x-533.79; 534.0x-534.79;<br>531.9x; 532.9x; 533.9x; 534.9x<br>Modified to remove:<br>531.00, 531.01, 531.20, 531.21,<br>531.40, 531.41, 531.60, 531.61<br>532.40, 532.41, 532.60, 532.61<br>533.40, 533.41, 533.60, 533.61,<br>534.00, 534.01, 534.20, 534.21,<br>534.40, 534.41, 534.60, 534.61 | K25, K26, K27, K28 | 1 |

| Condition | ICD-9 Code(s) | ICD-10 Code(s) | Point |
|---|---|---|---|
| Mild liver disease | 571.2x; 571.4x-571.69 | B18, K73, K74, K700, K701, K702,<br>K703, K709, K717, K713, K714, K715,<br>K760, K762, K763, K764, K768, K769,<br>Z944 | 1 |
| Diabetes (mild to moderate) | 250.0x-250.39, 250.7x | E100, E101, E106, E108, E109, E110,<br>E111, E116, E118, E119, E120, E121,<br>E126, E128, E129, E130, E131, E136,<br>E138, E139, E140, E141, E146, E148,<br>E149 | 1 |
| Diabetes + complications | 250.4x-250.69 | E102, E103, E104, E105, E107, E112,<br>E113, E114, E115, E117, E122, E123,<br>E124, E125, E127, E132, E133, E134,<br>E135, E137, E142, E143, E144, E145,<br>E147 | 2 |
| Hemiplegia or paraplegia | 342.xx; 344.1x | G81, G82, G041, G114, G801, G802,<br>G830, G831, G832, G833, G834, G839 | 2 |
| Renal disease | 582.xx; 583.0x-583.79; 585.xx-<br>586.99; 588.xx | N18, N19, N052, N053, N054, N055,<br>N056, N057, N250, I120, I131, N032,<br>N033, N034, N035, N036, N037, Z490,<br>Z491, Z492, Z940, Z992 | 2 |
| Any malignancy,<br>including<br>lymphoma and<br>leukemia | 140.xx-172.99; 174.xx-195.99;<br>200.xx-208.99 | C00, C01, C02, C03, C04, C05, C06, C07, C08, C09, C10, C11, C12, C13, C14, C15, C16, C17, C18, C19, C20, C21, C22, C23, C24, C25, C26, C30, C31, C32, C33, C34, C37, C38, C39, C40, C41, C43, C45, C46, C47, C48, C49, C50, C51, C52, C53, C54, C55, C56, C57, C58, C60, C61, C62, C63, C64, C65, C66, C67, C68, C69, C70, C71, C72, C73, C74, C75, C76, C81, C82, C83, C84, C85, C88, C90, C91, C92, C93, C94, C95, C96, C97 | 2 |
| Moderate/severe<br>liver disease | 456.0x-456.29; 572.2x-572.89<br>Modified to remove: 456.0x,<br>456.20 | K704, K711, K721, K729, K765, K766,<br>K767, I850, I859, I864, I982 | 3 |
| Metastatic solid tumor | 196.xx-199.99 | C77, C78, C79, C80 | 6 |
| AIDS | 042.xx-044.99 | B20, B21, B22, B24 | 6 |

**Table 11. Baseline Comorbidities** 

| Covariates | ICD-9-CM/CPT/HCPCS<br>Codes | ICD-10-CM Codes |
|---|---|---|
| History Stroke/SE | Same as the outcome<br>stroke/SE (Table 12) | Same as the outcome stroke/SE (Table 12) |
| History of Bleeding | Same as the outcome major bleeding (Table 12) | Same as the outcome major bleeding (Table 12) |
| Congestive Heart<br>Failure (CHF) | 398.91, 402.x1, 404.x3,<br>428.xx | I0981, I110, I132, I501, I5020, I5021, I5022, I5023, I5030, I5031, I5032, I5033, I5040, I5041, I5042, I5043, I509 |
| Diabetes | 250.xx, 357.2, 362.0, 366.41 | E08311, E08319, E083211, E083212, E083213, E083219, E083291, E083291, E083292, E083293, E083391, E083311, E083312, E083313, E083319, E083391, E083392, E083393, E083399, E083411, E083412, E083413, E083419, E083491, E083492, E083493, E083499, E083511, E083512, E083513, E083519, E083521, E083522, E083523, E083529, E083531, E083522, E083533, E083539, E083541, E083542, E083543, E083549, E083551, E083552, E083553, E083559, E083551, E083559, E083591, E083551, E083559, E083591, E083592, E083593, E083599, E0836, E0840, E0842, E09311, E09319, E093211, E093212, E093213, E093219, E093291, E093292, E093293, E093399, E093311, E093319, E093311, E093319, E093311, E093319, E093311, E093319, E093311, E093319, E093311, E093312, E093311, E093312, E093313, E093319, E093391, E093492, E093593, E093511, E093512, E093513, E093 |

| Covariates | ICD-9-CM/CPT/HCPCS<br>Codes | ICD-10-CM Codes |
|---|---|---|
| | | E113313, E113319, E113391, E113392, E113393, E113399, E113411, E113412, E113413, E113419, E113491, E113492, E113493, E113521, E113511, E113512, E113513, E113519, E113521, E113522, E113523, E113529, E113531, E113532, E113533, E113539, E113541, E113542, E113543, E113549, E113551, E113552, E113553, E113559, E113551, E113552, E113553, E113559, E113591, E113592, E113593, E113599, E1136, E1137X1, E1137X2, E1137X3, E1137X9, E1139, E1140, E1141, E1142, E1143, E1144, E1149, E1151, E1152, E1159, E11610, E11618, E11620, E11621, E11622, E11628, E11630, E11638, E11641, E11649, E1165, E1169, E118, E119, E1300, E1301, E1310, E1311, E1321, E1322, E1329, E13311, E13319, E133291, E133292, E133293, E133299, E13311, E133312, E133213, E133319, E133391, E133392, E133393, E133399, E133411, E133412, E133413, E133514, E133512, E133513, E133519, E133521, E133522, E133533, E133519, E133521, E133522, E133533, E133529, E133531, E133532, E1335349, E133532, E133539, E133539, E133541, E133542, E133543, E133549, E133552, E133553, E133559, E133559, E133551, E133522, E133553, E133559, E133551, E133522, E133551, E133522, E133553, E133559, E133641, E13649, E1365, E1369, E138, E139, E0851, E0852, E0951, E0952, E1051, E1052, E1151, E1152, E1351, E1352, E1359, E13610, E13618, E13620, E13618, E13660, E13618, E13620, E13618, E13620, E13638, E13641, E13649, E1365, E1369, E138, E1369, E138, E1399, E1386, E13630, E13638, E13641, E13649, E1365, E1369, E138, E1369, E138, E13600, E13618, E13620, E13618, E13620, E13621, E13622, E13628, E13630, E13638, E13641, E13649, E1365, E1369, E138, E1369, E138, E1399 |
| Hypertension | 401.xx -405.xx | I10, I110, I119, I120, I129, I130, I1310, I1311, I132, I150, I151, I152, I158, I159, I160, I161, I169, N262 |
| Renal Disease | 582.xx; 583.0x-583.79;<br>585.xx-586.99; 588.xx | B520, E0821, E0822, E0829, E0921, E0922, E0929, I120, I129, I130, I1310, I1311, I132, M3214, M3215, M3504, N000, N001, N002, N003, N004, N005, N006, N007, N008, N009, N010, N011, N012, N013, N014, N015, N016, N017, N018, N019, N020, N021, N022, N023, N024, N025, N026, N027, N028, N029, N030, N031, N032, N033, N034, N035, N036, N037, N038, N039, N040, N041, N042, N043, N044, N045, N046, N047, N048, N049, N050, N051, N052, N053, N054, N055, N056, N057, N058, N059, N060, N061, N062, N063, N064, N065, N066, |

| Covariates | ICD-9-CM/CPT/HCPCS<br>Codes | ICD-10-CM Codes |
|---|---|---|
| | | N067, N068, N069, N070, N071, N072, N073, N074, N075, N076, N077, N078, N079, N08, N140, N141, N142, N143, N144, N150, N158, N159, N16, N170, N171, N172, N178, N179, N181, N182, N183, N184, N185, N186, N189, N19, Z992, Z9115, Z4931, Z4901, Z4902, Z4931, Z4932, Z4932 Procedure codes: 5A1D00Z, 5A1D60Z, 05HY33Z, 06HY33Z, 03130ZD, 03140ZD, 03150ZD, 03160ZD, 03170ZD, 03180ZD, 03190ZF, 031209F, 03120AD, 03120AF, 03120JD, 03120JF, 03120F, 03120KD, 03120KF, 03120ZD, 03120ZF, 03130JD, 03130AF, 03130JF, 03130JF, 03130JF, 03130AD, 03130AF, 03130JF, 03130JF, 03140AD, 03140AF, 03140JD, 03140JF, 03140KD, 03140KF, 03140ZD, 03140ZF, 03150JD, 03150JF, 03150JF, 03150AD, 03150AF, 03150JD, 03150JF, 03150KD, 03150KF, 03150ZD, 03150ZF, 03160JD, 03160JF, 03160KD, 03160AF, 03160JD, 03160JF, 03160KD, 03160KF, 03160ZD, 03150ZF, 03170JF, 03170KD, 03170AD, 03170AF, 03170JD, 03170JF, 03170KD, 03170KF, 03170ZD, 03170ZF, 03180JD, 03180AF, 03180AF, 03180JF, 03180JF, 03180AF, 03180JF, 03180JF, 03180AF, 03180JF, 03180JF, 03180AF, 03180JF, 03180JF, 03180AF, 03180JF, 03180AF, 03180JF, 03180KD, 03180AF, 03180JF, 03180KF, 03190JF, 03180JF, 03190JF, 03190JF |
| Liver Disease | 570-573 | K70-K77 |
| Myocardial<br>Infarction | 410.xx, 412.xx | I2101, I2102, I2109, I2111, I2119, I2121, I2129, I213, I214, I220, I221, I222, I228, I229, I252 |
| Dyspepsia or | 787.1: Heartburn | |
| Stomach Discomfort | 789.0: Abdominal Pain | R100, R1010-R1012 |
| | 789.4: Abdominal Rigidity | |
| | 789.6: Abdominal Tenderness | |
| | 536.8: Dyspepsia | K30, R1013, R102, R10811, R10812, R10813,<br>R10814, R10816, R10817, R10819, R10821,<br>R10822, R10826, R10827, R10829, R1084, R109,<br>R12, R1930, R1931, R1932, R1936, R1937 |

| Covariates | ICD-9-CM/CPT/HCPCS<br>Codes | ICD-10-CM Codes |
|---|---|---|
| Peripheral artery disease | The state of the s | 1700, 1701, 170201, 170202, 170203, 170208, 170209, 170211, 170212, 170213, 170218, 170219, 170221, 170222, 170223, 170228, 170229, 170231, 170232, 170233, 170234, 170235, 170238, 170239, 170241, 170242, 170243, 170244, 170245, 170248, 170249, 17025, 170261, 170262, 170263, 170268, 170269, 170291, 170292, 170293, 170299, 170301, 170302, 170303, 170308, 170309, 170311, 170312, 170313, 170318, 170319, 170321, 170322, 170323, 170338, 170338, 170339, 170331, 170332, 170333, 170334, 170335, 170338, 170339, 170341, 170342, 170343, 170344, 170345, 170368, 170369, 170391, 170392, 170393, 170398, 170399, 170401, 170402, 170403, 170408, 170409, 170411, 170412, 170413, 170418, 170419, 170421, 170422, 170423, 170428, 170438, 170439, 170441, 170442, 170443, 170444, 170445, 170448, 170449, 170471, 170401, 170402, 170403, 170408, 170409, 170411, 170401, 170402, 170403, 170438, 170439, 170391, 170392, 170393, 170493, 170449, 170421, 170442, 170443, 170448, 170445, 170449, 170451, 170462, 170463, 170468, 170469, 170491, 170492, 170493, 170498, 170499, 170501, 170502, 170503, 170508, 170509, 170511, 170512, 170513, 170518, 170519, 170521, 170522, 170523, 170528, 170529, 170531, 170532, 170533, 170534, 170544, 170544, 170545, 170566, 170566, 170567, 170567, 170567, 170568, 170569, 170591, 170593, 170598, 170599, 170601, 170602, 170603, 170608, 170609, 170611, 170612, 170613, 170618, 170619, 170621, 170622, 170633, 170638, 170639, 170641, 170642, 170663, 170668, 170669, 170691, 170692, 170693, 170799, 170711, 170712, 170713, 170718, 170719, 170721, 170722, 170723, 170728, 170738, 170799, 170711, 170712, 170713, 170718, 170719, 170721, 170722, 170723, 170728, 170738, 170739, 170741, 170742, 170743, 170744, 170745, 170744, 170747, 170799, 170791, 170792, 170793, 170798, 170799, 170711, 170792, 170793, 170798, 170799, 170711, 170772, 170773, 170774, 170777, 170779, 17071, 17079, 17091, 17092, 17000, 17011, 1 |

| Covariates | ICD-9-CM/CPT/HCPCS<br>Codes | ICD-10-CM Codes |
|---|---|---|
| Non-stroke/SE<br>peripheral vascular<br>disease | 440, 441, 442, 443 | 170-173, 177-179 |
| Transient ischemic attack (TIA) | 435.x | G458, G459, Z8673 |
| Coronary artery disease | 410.xx-414.xx | I200, I201, I208, I209, I2101, I2102, I2109, I2111, I2119, I2121, I2129, I213, I214, I220, I221, I222, I228, I229, I240, I241, I248, I249, I2510, I25110, I25111, I25118, I25119, I252, I253, I2541, I2542, I255, I256, I25700, I25701, I25708, I25709, I25710, I25711, I25718, I25719, I25720, I25721, I25728, I25729, I25730, I25731, I25738, I25739, I25750, I25751, I25758, I25759, I25760, I25761, I25768, I25769, I25790, I25791, I25798, I25799, I25810, I25811, I25812, I2582, I2583, I2584, I2589, I259 |
| Anemia and coagulation defects | 280.xx-286.xx | D50-D53, D55-D59, D60-D69, |

Table 12. Clinical Outcomes

| Outcome Variables | | ICD-9-CM/Procedure<br>Codes | ICD-10-CM Codes/Procedure Codes |
|---|---|---|---|
| Stoke/<br>SE | Hemorrhagic<br>Stroke | 430.xx-432.xx Cases will<br>be excluded if traumatic<br>brain injury (ICD-9:<br>800-804, 850-854) was<br>present during<br>hospitalization. | I6000, I6001, I6002, I6010, I6011, I6012, I602, I6030, I6031, I6032, I604, I6050, I6051, I6052, I606, I607, I608, I609, I610, I611, I612, I613, I614, I615, I616, I618, I619; Cases will be excluded according to Table 12. |
| | Ischemic<br>Stroke | 433.x1, 434.x1, 436 | I6300, I63011, I63012, I63013, I63019, I6302, I63031, I63032, I63033, I63039, I6309, I6310, I63111, I63112, I63113, I63119, I6312, I63131, I63132, I63133, I63139, I6319, I6320, I63211, I63212, I63213, I63219, I6322, I63231, I63232, I63233, I63239, I6329, I6330, I63311, I63312, I63313, I63319, I63321, I63322, I63323, I63329, I63331, I63332, I63339, I63339, I63341, I63342, I63343, I63349, I6339, I6340, I63411, I63412, I63413, I63419, I63421, I63422, I63423, I63429, I63431, I63432, I63439, I63439, I63441, I63442, I63443, I63449, I6349, I6350, I63511, I63512, I63513, I63519, I63521, I63522, I63523, I63529, I63531, I63532, I63539, I63541, I63542, I63543, I63549, I6359, I636, I638, I639, I6789 |
| | Systemic | 444.x, 445.x | I7401, I7409, I7410, I7411, I7419, I742, I743, |

| Outco | ome Variables | ICD-9-CM/Procedure<br>Codes | ICD-10-CM Codes/Procedure Codes |
|---|---|---|---|
| | Embolism | | I744, I745, I748, I749, I75011, I75012, I75013, I75019, I75021, I75022, I75023, I75029, I7581, I7589 |
| Major<br>Bleedi<br>ng | Major<br>Gastrointestinal<br>bleeding event | 456.0, 456.20, 530.82,<br>531.0x, 531.2x, 531.4x,<br>531.6x, 532.0x, 532.2x,<br>532.4x, 532.6x, 533.0x,<br>533.2x, 533.4x, 533.6x,<br>534.0x, 534.2x, 534.4x,<br>534.6x, 535.01, 535.11,<br>535.21, 535.31, 535.41,<br>535.51, 535.61, 537.83,<br>562.02, 562.03, 562.12,<br>562.13, 568.81, 569.3,<br>569.85, 578.x;<br>Procedure Code: 44.43 | I8501, I8511, K2211, K226, K250, K252, K254, K256, K260, K262, K264, K266, K270, K272, K274, K276, K280, K282, K284, K286, K2901, K2921, K2931, K2941, K2951, K2961, K2971, K2981, K2991, K31811, K3182, K5521, K5701, K5711, K5713, K5721, K5731, K5733, K5741, K5751, K5753, K5781, K5791, K5793, K625, K6381, K661, K920, K921, K922, K9161, K9162, K91840, K91841 |
| | Major<br>Intracranial<br>Hemorrhage<br>(ICH) | 430, 431, 432.0, 432.1,<br>432.9, 852.0x, 852.2x,<br>852.4x, 853.0x | I6000, I6001, I6002, I6010, I6011, I6012, I602, I6030, I6031, I6032, I604, I6050, I6051, I6052, I606, I607, I608, I609, I610, I611, I612, I613, I614, I615, I616, I618, I619, I6200, I6201, I6202, I6203, I621, I629, S06340A, S06341A, S06342A, S06343A, S06344A, S06345A, S06346A, S06347A, S06348A, S06349A, S06350A, S06351A, S06352A, S06353A, S06354A, S06355A, S06356A, S06357A, S06358A, S06359A, S06360A, S06361A, S06362A, S06363A, S06364A, S06363A, S06364A, S06363A, S06364A, S06365A, S06367A, S06368A, S06369A, S064X0A, S064X1A, S064X2A, S064X3A, S064X4A, S064X5A, S065X0A, S065X1A, S065X2A, S065X3A, S065X4A, S065X3A, S065X4A, S065X5A, S066X0A, S066X1A, S066X2A, S066X3A, S066X4A, S066X5A, S066X6A, S066X5A, S066X6A, S066X7A, S066X8A, S066X9A |
| | Major Other<br>hemorrhage | 285.1, 360.43, 362.43,<br>362.81, 363.61, 363.62,<br>363.72, 364.41, 372.72,<br>374.81, 376.32, 377.42,<br>379.23, 423.0x, 596.7x,<br>599.7x, 602.1x, 620.1,<br>621.4, 626.2, 626.5, 626.7,<br>626.8, 626.9, 719.1x,<br>782.7, 784.7, 784.8,<br>786.3x, 958.2, 997.02,<br>998.11;<br>Procedure codes: 99.04 | D62, D7801, D7802, D7821, D7822, E3601, E3602, E89810, E89811, G9731, G9732, G9751, G9752, H05231, H05232, H05233, H05239, H1130, H1131, H1132, H1133, H2100, H2101, H2102, H2103, H31301, H31302, H31303, H31309, H31311, H31312, H31313, H31319, H31411, H31412, H31413, H31419, H3560, H3561, H3562, H3563, H35731, H35732, H35733, H35739, H4310, H4311, H4312, H44313, H44811, H44812, H44813, H44819, H47021, H47022, H47023, H47029, H59111, H59112, H59113, H59119, H59121, H59122, H59123, H59129, H59311, H59312, H59313, H59319, |

| Outcome Variables | ICD-9-CM/Procedure<br>Codes | ICD-10-CM Codes/Procedure Codes |
|---|---|---|
| | | H59321, H59322, H59323, H59329, H9521, H9522, H9541, H9542, I312, I97410, I97411, I97418, I9742, I97610, I97611, I97618, I97620, J9561, J9562, J95830, J95831, L7601, L7602, L7621, L7622, M2500, M25011, M25012, M25019, M25021, M25022, M25029, M25031, M25032, M25039, M25041, M25042, M25049, M25051, M25052, M25059, M25061, M25062, M25069, M25071, M25072, M25073, M25074, M25075, M25076, M2508, M96810, M96811, M96830, M96831, N421, N857, N897, N920, N923, N930, N938, N939, N9961, N9962, N99820, N99821, R040, R041, R042, R0489, R049, R233, R310, R319, R58, T792XXA; Procedure codes: 30230N1, 30230P1, 30233N1, 30233P1, 30240N1, 30240P1, 30243N1, 30243P1, 30250N1, 30260P1, 30263N1, 30263P1 |